## **Document Coversheet**

Study Title: Interactions of Alcohol and Opioids: Pharmacodynamic Effects

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 9/2/2025 |
| NCT Number: | NCT04300751 |
| IRB Number | 55176 |
| Coversheet created: | 10/13/2025 |

0 ι

IRB Approval 9/2/2025 IRB # 55176 IRB2

#### **IMPORTANT NOTE:**

If you accidentally select the wrong IRB type or "Protocol Process Type" while your Initial Review (IR) application is in draft form (unsubmitted), you may change your selections. Please contact the Office of Research Integrity (ORI) at 859-257-9428, <a href="mailto:IRBsubmission@uky.edu">IRBsubmission@uky.edu</a>, or request a consult to resolve any questions regarding your selections *prior* to submitting your Initial Review application.

If your submitted IR application has been returned to you for requested revisions or additional information, to streamline the review process do not make changes to your selections here unless instructed to do so by the ORI/IRB.

Changes to this section cannot be made after initial approval has been issued (the option is not available for MR or CR).

For guidance, see:

- Which IRB should review my research?
- Which Protocol Process Type?
- "Getting Started"

| Which IRB @ Medical @ NonMedical |
|---|
| Protocol Process Type © Exemption © Expedited (Must be risk level 1) © Full |

The revised Common Rule expanded exemption certification category 4 for certain secondary research with identifiable information or biospecimens. The regulations no longer require the information or biospecimens to be existing. For more information see the Exemption Categories Tool.

## **EXPEDITED CERTIFICATION**

0 unresolved comment(s)

#### To Be Completed Only If Protocol is to Receive Expedited Review

#### **Applicability**

- A. Research activities that (1) present no more than \*minimal risk to human subjects, and (2) involve only procedures listed in one or more of the following categories, may be reviewed by the IRB through the expedited review procedure authorized by 45 CFR 46.110 and 21 CFR 56.110. The activities listed should not be deemed to be of minimal risk simply because they are included on this list. Inclusion on this list merely means that the activity is eligible for review through the expedited review procedure when the specific circumstances of the proposed research involve no more than minimal risk to human subjects.
- B. The categories in this list apply regardless of the age of subjects, except as noted.
- C. The expedited review procedure may not be used where identification of the subjects and/or their responses would reasonably place them at risk of criminal or civil liability or be damaging to the subjects' financial standing, employability, insurability, reputation, or be stigmatizing, unless reasonable and appropriate protections will be implemented so that risks related to invasion of privacy and breach of confidentiality are no greater than minimal.
- D. The expedited review procedure may not be used for classified research involving human subjects.
- E. IRBs are reminded that the standard requirements for informed consent (or its waiver, alteration, or exception) apply regardless of the type of review—expedited or convened—utilized by the IRB.
  - \*"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves from those ordinarily encountered in daily life or during the performance of routine physical or psychological examination or tests. 45 CFR 46.102(i)

Check the appropriate categories that apply to your research project:

- ✓ Study was originally approved by the full IRB at a convened meeting.
- □1) Clinical studies of drugs and medical devices only when condition (a) or (b) is met.
  - A. Research on drugs for which an investigational new drug application is not required. (Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)
  - B. Research on medical devices for which (i) an investigational device exemption application is not required\*; or (ii) the medical device is cleared/approved for marketing and the medical device is being used in accordance with its cleared/approved labeling.\*\*
  - \* Study must meet one of the IDE Exempt categories listed on the Device Form Attachment.
  - \*\* An approved Device used in research according to its approved labeling is considered Exempt from IDE requirements. NOTE: Select Category 1 for compassionate use medical device applications or individual patient expanded access investigational drug applications for which FDA has waived the requirement for full review.
- □2) Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture as follows:
  - A. From healthy, nonpregnant adults who weigh at least 110 pounds. For these subjects, the amounts drawn may not exceed 550 ml in an 8 week period and collection may not occur more frequently than 2 times per week; or
  - B. From other adults and children\* considering the age, weight, and health of the subjects, the collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period and collection may not occur more frequently than 2 times per week.

NOTE: Intravenous (IV), Port, Central, or any other lines are NOT eligible under this category even if the research involves "minimal risk".

\*In Kentucky, "child/children" refers to all individuals less than 18 years of age unless the individual(s) is/are legally emancipated. (See Informed Consent SOP for discussion of "Emancipated Individuals" under Kentucky state law.) Individuals less than 18 years of age who are not emancipated meet the federal definition for "child" (e.g., DHHS, FDA, and U.S. Department of Education). Children are defined in the HHS regulations as "persons who have not attained the legal age for consent to treatments or procedures involved in the research, under the applicable law of the jurisdiction in which the research will be conducted." If conducting research outside the state of Kentucky, you are responsible for complying with applicable state law.

□ 3) Prospective collection of biological specimens for research purposes by noninvasive means. Examples:

- A. Hair and nail clippings in a nondisfiguring manner;
- B. Deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction;
- C. Permanent teeth if routine patient care indicates a need for extraction;
- D. Excreta and external secretions (including sweat);
- E. Uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gumbase or wax or by applying a dilute citric solution to the tongue;
- F. placenta removed at delivery;
- G. Amniotic fluid obtained at the time of rupture of the membrane prior to or during labor;
- H. Supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic scaling of the teeth and the process is accomplished in accordance with accepted prophylactic techniques;
- I. Mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings;
- J. Sputum collected after saline mist nebulization.
- □4) Collection of data through noninvasive procedures (not involving general anesthesia or sedation) routinely employed in clinical practice, excluding procedures involving x-rays or microwaves. Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, including studies of cleared medical devices for new indications.) Examples:
  - A. Physical sensors that are applied either to the surface of the body or at a distance and do not involve input of significant amounts of energy into the subject or an invasion of the subject's privacy;
  - B. Weighing or testing sensory acuity;
  - C. Magnetic resonance imaging;
  - D. electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, doppler blood flow, and echocardiography;
  - E. moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the age, weight, and health of the individual.
- □5) Research involving materials (data, documents, records, or specimens) that have been or will be collected solely for non-research purposes (such as medical treatment or diagnosis) as well as research involving existing information or specimens that were previously collected for research purposes, provided they were not collected for the currently proposed research. (Note: Some research in this category may qualify for Exempt review. This listing refers only to research that is not exempt.) (Note: If submission includes materials previously collected for either non-research or research purposes in a protocol for which IRB approval expired, you may check Category 5. However, a separate category must also be selected for prospective collection of data/specimens obtained solely for research purposes)
- □ 6) Collection of data from voice, video, digital, or image recordings made for research purposes.
- □7) Research on individual or group characteristics or behavior (including, but not limited to, research on perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (Note: Some research in this category may be exempt from the HHS regulations for the protection of human subjects. This listing refers only to research that is not exempt.)

#### **CONTINUATION REVIEW/FINAL REVIEW**

0 unresolved comment(s)

In accordance with federal regulations and/or local policies, the IRB conducts periodic review of all currently approved projects. If you need your IRB approval to continue and you do not complete and submit the required materials in a timely manner, IRB approval will expire at the end of your current approval period.

If you have any questions, please contact the Office of Research Integrity at 859-257-9428 or email IRBsubmission@uky.edu.

To initiate your continuation review (CR)/annual administrative review (AAR), or properly close your study, complete this section and update/correct all other sections of your IRB application as applicable.

\*\*\*IMPORTANT\*\*\* Before leaving this page to update other sections of your application, be sure to SAVE this section first.



#### 1. Status of the Research

Check the statement(s) that best describe(s) the current status of your research: 0

- □ No subjects have enrolled to date.
- □ Recruitment and/or enrollment of new subjects or review of records/specimens continue.
- ☐ Study is closed to enrollment, but subjects still receive research-related interventions (e.g., treatment, blood draws).
- □ Study enrollment is permanently closed; subjects have completed all research-related interventions; and the study remains active only for long-term follow-up of subjects (see Tool Tip above for info on long-term follow-up of subjects).\*
- □ Research has progressed to the point that it involves 1) Data analysis, including analysis of identifiable private information or identifiable biospecimens; and/or 2) Accessing follow-up clinical data from procedures that subjects would undergo as part of clinical care.\*
- □ The remaining research activities are limited only to data analysis. There is no subject/record/specimen identifying codes or links to the data; the researcher or research team cannot readily ascertain the subject's identity.\*
- ☐ All study activities are complete. IRB approval can be inactivated.
- \*Possibility that review will move from Full to Expedited.

## 2. If subjects have been enrolled within the last year, and the IRB approved a consent/assent form for your study:

Please attach a complete, signed copy for the last two subjects enrolled with **each** consent/assent form/HIPAA form since the last annual review.

(Example: If 3 different approved consent forms were used since the last annual review, please provide the two most recent signed copies of each version for a total of six.)

#### Attachments

| Attach Type | File Name |
|---|---|
| Entire Signed Consent Form | Signed Consents - 1 Screening & 1 Main Study.pdf |

#### 3. Informed Consent

If the study is open to subject enrollment, please go to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- One clean copy in PDF (without the IRB Approval stamp) of the currently approved consent/assent document(s), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is open to subject enrollment and the IRB has waived the requirement to document informed consent, please go to the Informed Consent section of the E-IRB Application and verify attachment(s) include:

- One clean copy in PDF of the currently approved document used for the informed consent process (e.g., cover letter, phone script), or,
- If requesting changes to the consent/assent document(s), submit one copy with the changes highlighted (and designate Document Type as "Highlighted"), and one clean copy in PDF (without the changes highlighted).

If the study is closed to subject enrollment, please go to the Informed Consent section of the E-IRB Application and remove Informed Consent Documents designated to get an IRB approval stamp to avoid having them appear valid for enrollment.

## 4. Unanticipated Problems Involving Risk to Subjects or Others/Adverse Events Summary & Assessment

Did any problems/adverse events occur during the last 12 months?

Yes ○ No

In the space below, provide a written summary of both unanticipated problems\* and available information regarding adverse events since the last review (e.g., initial review or annual/continuing review). The amount of detail provided in such a summary will vary depending on the type of research being conducted; in many cases, such a summary could be a brief statement that there have been no unanticipated problems and that adverse events have occurred at the expected frequency and level of severity as documented in the research protocol, the informed consent document, and investigator's brochure (if applicable). The summary must include the Pl's assessment whether the problems/adverse events warrant changes to the protocol, consent process, or risk/benefit ratio.

Note: It is the IRB's expectation that all unanticipated problems involving risk to subjects or others or related deaths requiring prompt reporting are submitted in the appropriate time frame (See Policy [PDF]). Your response to this Annual/Continuing Review is considered assurance that all prompt reportable problems/adverse events have been submitted for IRB review.

Since the last continuation review, there have been NO adverse events. There have been a total of 10 adverse events since study initiation; all resolved without sequelae. These AEs did not warrant any changes to the protocol, consent process, or risk/benefit ratio. Since study initiation, there have been no serious adverse events.

\*For multisite studies, the written summary should describe external events determined to be unanticipated problems involving risk to subjects or others.

| 5. Subject Info To-Date |
|---|
| Our records for the previously approved IRB application indicate the <b>IRB approved estimate</b> of subjects to be enrolled (or records/specimens reviewed) is: |
| Enter the number of enrolled subjects (or records/specimens reviewed) that have not been previously reported to the IRB |
| Our records for the previously approved IRB application indicate the previous total # of subjects enrolled (or records/specimens reviewed) since activation of the study is: |
| The new total number of subjects enrolled (or records/specimens reviewed) since activation of the study: 24 |
| Please review the Project Info section for the IRB approved estimate of subjects to be enrolled (or records/specimens reviewed). If this new total exceeds your approved estimate of subjects to be enrolled (or records/specimens reviewed), please update the number in the field for Number of Human Subjects in the Project Info section. |

## 6. Data and Safety Monitoring Board (DSMB)/Plan (DSMP)

If your study is monitored by a DSMB or under a DSMP, attach all documentation (i.e. summary report; meeting minutes) representing Data and Safety Monitoring activities that have not been previously reported to the IRB.

Attachments

## 7. Since the most recent IRB Initial/Continuation Review Approval:

Have there been any participant complaints regarding the research?

associated with the research?

| | 55176 |
|---|---|
| ∩ Yes ∈ No | |
| If yes, in the field below, provide a summary describing the complaints. | |
| Have any <b>subjects withdrawn</b> from the research voluntarily or by you as the PI for reasons related to safety, we lated to the conduct of the research? If a participant does not meet the screening criteria for a study even if the consent it is NOT considered a withdrawal. | |
| ⊂Yes ∈ No | |
| If yes, in the field below, provide a detailed explanation to the withdrawal(s) including if participants were lost to | contact. |
| Has any <b>new and relevant literature</b> been published since the last IRB review, especially literature relating | to risks associated wi<br>the research |
| If yes, attach a copy of the literature as well as a brief summary of the literature including, if pertinent, the impact protection of human subjects. | t of the findings on the |
| Attachments | |
| Have there been any interim findings? | |
| ⊂Yes ∈ No | |
| If yes, attach a copy of Interim Findings. | |
| Attachments | |

## Have subjects experienced any benefits?

If yes, in the field below, provide a description of benefits subjects have experienced.

Have there been any inspections/audits/quality improvement reviews of your research protocol resulting in the need for corrective action in order to protect the safety and welfare of subjects?

If yes, please attach documentation evidencing the outcome(s) and any corrective action(s) taken as a result.

## Attachments

Was an FDA 483 issued as a result of any inspections/audits?

If yes, submit documentation using attachment button above.

#### 8. Risk Level:

Our records for the previously approved IRB application show your research is:

Risk Level: 3

Has something during the course of your research changed the level of risk?

Yes ○ No

If yes, go to the Risk Level section, mark the appropriate risk level, and in the field below, describe why the risk level has changed:

Protocol closed to enrollment; open for data analysis only.

## 9. Funding/Support:

Our records for the **previously approved IRB** application indicate your research is being submitted to, supported by, or conducted in cooperation with the following external or internal agency(ies) or funding program(s):

| | l | □ Grant application pending |
|---|---|---|
| ☐ (CDC) Centers for Disease Control & Prevention ☐ (HRSA) Health Resources and Services Administration ☐ (SAMHSA) Substance Abuse and Mental Health Services Administration ☐ (DoJ) Department of Justice or Bureau of Prisons ☐ (DoE) Department of Energy ☐ (EPA) Environmental Protection Agency ☐ Federal Agencies Other Than Those Listed Here ☐ Industry (Other than Pharmaceutical Companies) ☐ Internal Grant Program w/ proposal ☐ Internal Grant Program w/o proposal ☐ National Science Foundation ☐ Other Institutions of Higher Education ☐ Pharmaceutical Company ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | Œ (HHS) Dept. of Health & Human Services |
| ■ (HRSA) Health Resources and Services Administration ■ (SAMHSA) Substance Abuse and Mental Health Services Administration ■ (DoJ) Department of Justice or Bureau of Prisons ■ (DoE) Department of Energy ■ (EPA) Environmental Protection Agency ■ Federal Agencies Other Than Those Listed Here ■ Industry (Other than Pharmaceutical Companies) ■ Internal Grant Program w/ proposal ■ Internal Grant Program w/o proposal ■ National Science Foundation ■ Other Institutions of Higher Education ■ Pharmaceutical Company ■ Private Foundation/Association ■ U.S. Department of Education ■ State | l | ✓ (NIH) National Institutes of Health |
| ☐ (SAMHSA) Substance Abuse and Mental Health Services Administration ☐ (DoJ) Department of Justice or Bureau of Prisons ☐ (DoE) Department of Energy ☐ (EPA) Environmental Protection Agency ☐ Federal Agencies Other Than Those Listed Here ☐ Industry (Other than Pharmaceutical Companies) ☐ Internal Grant Program w/ proposal ☐ Internal Grant Program w/o proposal ☐ National Science Foundation ☐ Other Institutions of Higher Education ☐ Pharmaceutical Company ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | □ (CDC) Centers for Disease Control & Prevention |
| <ul> <li>□ (DoJ) Department of Justice or Bureau of Prisons</li> <li>□ (DoE) Department of Energy</li> <li>□ (EPA) Environmental Protection Agency</li> <li>□ Federal Agencies Other Than Those Listed Here</li> <li>□ Industry (Other than Pharmaceutical Companies)</li> <li>□ Internal Grant Program w/ proposal</li> <li>□ Internal Grant Program w/o proposal</li> <li>□ National Science Foundation</li> <li>□ Other Institutions of Higher Education</li> <li>□ Pharmaceutical Company</li> <li>□ Private Foundation/Association</li> <li>□ U.S. Department of Education</li> <li>□ State</li> </ul> | l | |
| □ (DoE) Department of Energy □ (EPA) Environmental Protection Agency □ Federal Agencies Other Than Those Listed Here □ Industry (Other than Pharmaceutical Companies) □ Internal Grant Program w/ proposal □ Internal Grant Program w/o proposal □ National Science Foundation □ Other Institutions of Higher Education □ Pharmaceutical Company □ Private Foundation/Association □ U.S. Department of Education □ State | l | |
| ☐ (EPA) Environmental Protection Agency ☐ Federal Agencies Other Than Those Listed Here ☐ Industry (Other than Pharmaceutical Companies) ☐ Internal Grant Program w/ proposal ☐ Internal Grant Program w/o proposal ☐ National Science Foundation ☐ Other Institutions of Higher Education ☐ Pharmaceutical Company ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | □ (DoJ) Department of Justice or Bureau of Prisons |
| ■ Federal Agencies Other Than Those Listed Here ■ Industry (Other than Pharmaceutical Companies) ■ Internal Grant Program w/ proposal ■ Internal Grant Program w/o proposal ■ National Science Foundation ■ Other Institutions of Higher Education ■ Pharmaceutical Company ■ Private Foundation/Association ■ U.S. Department of Education ■ State | l | □ (DoE) Department of Energy |
| <ul> <li>☐ Industry (Other than Pharmaceutical Companies)</li> <li>☐ Internal Grant Program w/ proposal</li> <li>☐ Internal Grant Program w/o proposal</li> <li>☐ National Science Foundation</li> <li>☐ Other Institutions of Higher Education</li> <li>☐ Pharmaceutical Company</li> <li>☐ Private Foundation/Association</li> <li>☐ U.S. Department of Education</li> <li>☐ State</li> </ul> | l | □ (EPA) Environmental Protection Agency |
| ☐ Internal Grant Program w/ proposal ☐ Internal Grant Program w/o proposal ☐ National Science Foundation ☐ Other Institutions of Higher Education ☐ Pharmaceutical Company ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | ⊏ Federal Agencies Other Than Those Listed Here |
| <ul> <li>Internal Grant Program w/o proposal</li> <li>National Science Foundation</li> <li>Other Institutions of Higher Education</li> <li>Pharmaceutical Company</li> <li>Private Foundation/Association</li> <li>U.S. Department of Education</li> <li>State</li> </ul> | l | □ Industry (Other than Pharmaceutical Companies) |
| ■ National Science Foundation ■ Other Institutions of Higher Education ■ Pharmaceutical Company ■ Private Foundation/Association ■ U.S. Department of Education ■ State | l | ⊏ Internal Grant Program w/ proposal |
| □ Other Institutions of Higher Education □ Pharmaceutical Company □ Private Foundation/Association □ U.S. Department of Education □ State | l | ⊏Internal Grant Program w/o proposal |
| ☐ Pharmaceutical Company ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | □ National Science Foundation |
| ☐ Private Foundation/Association ☐ U.S. Department of Education ☐ State | l | □ Other Institutions of Higher Education |
| ■ U.S. Department of Education ■ State | l | □ Pharmaceutical Company |
| □ State | l | □ Private Foundation/Association |
| | l | □ U.S. Department of Education |
| Other: | l | □ State |
| | | Other: |
| | l | |

Please **update the Funding/Support section of your IRB application** if needed, including the following attachments if they contain changes not previously reported to the IRB:

- A current copy of your protocol if you are conducting industry/pharmaceutical research;
- A current Investigator Brochure (submit a copy with all changes underlined).
- A new or revised grant application for this project.

Did your project receive extramural funding?

Yes ○ No

If yes, please review and correct if necessary, the OSPA Account # information under the **Funding/Support section** of your IRB application.

If the project is externally funded, has the sponsor offered any of the research team enrollment incentives or other personal benefit bonuses? (e.g., cash/check, travel reimbursements, gift checks, etc.)

○Yes ○No ○N/A

Note: It is University of Kentucky policy that personal benefit bonuses are not allowed. If these conditions change during the course of the study, please notify the IRB.

## 10. Project Information

Our records for the previously approved IRB application indicate your estimated project end date is:

## 06/30/2026

If you have a new estimated project end date, please go to the Project Info section and change the date in the field for Anticipated Ending Date of Research Project.

## 11. Study Personnel

Our records for the previously approved IRB application indicate the following individuals are study personnel on this project (if applicable):

| Last Name | First Name |
|-----------|------------|
| Andrews | Lelia |

| Last Name | First Name |
|---------------|------------|
| Babalonis | Shanna |
| Canedo | Anabel |
| Christian | Eli |
| Dowden-Kruger | Melinda |
| Fanucchi | Laura |
| Fuller | Grayson |
| Hash | Matthew |
| Hunt | Cassandra |
| Lofwall | Michelle |
| Murphy | John |
| Nuzzo | Paul |
| Perpar | Justin |
| Randolph | Carly |
| Stafford | Maribeth |
| VanMeter | Connor |
| Vessels | Victoria |

Please review the individuals listed above and update your records as needed in the Study Personnel section of the E-IRB application, being sure that each individual listed has completed or is up-to-date on the mandatory human research protection training [see the policy on <u>Mandatory Human Subject Protection Training FAQs</u> (required every three years)].

## 12. Progress of the Research

To meet federal requirements the IRB is relying on your RESEARCH DESCRIPTION as a protocol summary and their expectation is that it is up-to-date. If the currently approved protocol (or research description) in your E-IRB application is outdated, please make applicable changes, and describe in the field below any substantive changes and explain why they are essential. If none, insert "N/A" in the text field below. If you are closing your study, you may use the space below to summarize the final status of the research.

N/A - See attached Progress Reported dated 18AUG2025.

Note: No changes in the research procedures should have occurred without previous IRB review. Approval from the IRB must be obtained before implementing any changes.

Provide a brief **summary** of any **modifications that affect subject safety and/or welfare** approved by the IRB since the last initial or continuation review (If none, insert "N/A" in the text field below.):

N/A - See attached Progress Reported dated 18AUG2025.

Attach one copy of the most recent progress report sent to the FDA, if available. All PI-sponsored IND/IDE studies are required to submit a copy of the FDA progress report.

Attachments

#### 13. Confidentiality/Security

Review your Research Description section and update the Confidentiality portion, if necessary, to describe measures for security of

## 14. Subject Demographics

Our records for the previously approved IRB application indicate the following categories of subjects and controls are included in your research:

- ☐ Children (individuals under age 18)
- Wards of the State (Children)
- Emancipated Minors
- Students
- **■** College of Medicine Students
- **UK Medical Center Residents or**

**House Officers** 

- Impaired Consent Capacity Adults
- Pregnant Women/Neonates/Fetal

Material

- □ Prisoners
- Non-English Speaking
- International Citizens
- Normal Volunteers
- Military Personnel and/or DoD

Civilian Employees

- □ Patients
- Appalachian Population

Please review the Subject Demographics section of your IRB application for accuracy, and note the following:

If during the course of your research 1) any prisoners have been enrolled, OR 2) subjects have been enrolled that became involuntarily confined/detained in a penal institution that have not been previously reported to the IRB, go to Subject Demographic section in your E-IRB application and mark "prisoners" in the categories of subjects to be included in the study, if it is not already marked.

Note: If either 1 or 2 above apply, and you have received funding from the Department of Health and Human Services (HHS), a Certification Letter should have been submitted to the Office for Human Research Protections (OHRP); prisoners and individuals who have become involuntarily confined/detained in a penal institution cannot continue participation in the research until OHRP issues approval. If the Certification has not been submitted, contact the Office of Research Integrity.

Based on the total # of subjects who have enrolled, complete the subject demographic section below:

| | Participant Demographics | | | |
|---|---|---|---|---|
| | Cisgender Man 🕕 | Cisgender Woman 🛈 | TGNB/TGE 🕕 | Unknown/Not Reported |
| American | | | | |
| Indian/Alaskan | | | | |
| Native | | | | |
| Asian | | | | |
| Black or | | | | |
| African | 4 | 2 | | |
| American | | | | |
| Latinx | 1 | | | |
| Native | | | | |
| Hawaiian or | | | | |
| Other Pacific | | | | |
| Islander | | | | |
| White | 17 | | | |
| American | | | | |
| Arab/Middle | | | | |
| Eastern/North | | | | |
| African | | | | |

| | <br>331 | 70 |
|----------------|---------|----|
| Indigenous | | |
| People | | |
| Around the | | |
| Wor <b>l</b> d | | |
| More than | | |
| One Race | | |
| Unknown or | | |
| Not Reported | | |

If unknown, please explain why:

Participant demographic information collected using NIH reporting format. Demographic information was not collected on cis/transgender status or the newly established race/ethnicity categories. Therefore, participants are reported as cisgender as none reported taking hormone therapies or having completed gender reassignment surgery at screening (although we acknowledge it is possible that an individual may identify as transgender without these interventions, cisgender seems to be the most appropriate designation). Furthermore, participants previously reported as "Mixed Race/Other" are now reported in the "More than One Race" category.

#### 15. Research Sites

Our records for the previously approved IRB application indicate that you are conducting research at the following sites:

■ UK Classroom(s)/Lab(s)
■ UK Clinics in Lexington
■ UK Clinics outside of Lexington
■ UK Healthcare Good Samaritan Hospital
■ UK Hospital

Schools/Education Institutions Schools/Education

Institutions

■ Fayette Co. School Systems \*

■ Other State/Regional School Systems

■ Institutions of Higher Education (other than UK)

Other Medical Facilities

■ Bluegrass Regional Mental Health Retardation Board

□ Cardinal Hill Hospital

■ Eastern State Hospital

■ Nursing Homes

■ Shriner's Children's Hospital

■ Other Hospitals and Med. Centers

■ Correctional Facilities

■ Home Health Agencies

■ International Sites

Other:

UK Robert Straus Research Building

If the above listed sites are not accurate, go to the Research Sites section of the E-IRB application to update the facilities at which research procedures have been or will be conducted.

If you are adding a new off-site facility, you may also need to update your E-IRB application Research Description, Research Sites, Informed Consent, and other affected sections as well as any documents which will list the off-site facility. Documents needing updating may include, but not limited to:

- Consent forms (attachment under Informed Consent section)
- Brochures (attachment under Additional Info section)
- Advertisements (attachment under Research Description section);
- Letter of support (attachment under Research Sites section)).

Please revise applicable sections and attachments as necessary.

## 16. Disclosure of Significant Financial Interest

Disclosure of Significant Financial Interest:

Our records for the previously approved IRB application indicate that you, your investigators, and/or key personnel (KP) have a significant financial interest (SFI) related to your/their responsibilities at the University of Kentucky (that requires disclosure per the UK administrative regulation 7:2): 1

If you need to update your records, please go to the PI Contact Information section and/or Details for individuals listed in the Study Personnel section to change your response to the applicable question(s).

## 17. Supplementals

To ensure the IRB has the most accurate information for your protocol you are expected to re-visit the E-IRB application sections and make corrections or updates as needed. At a minimum you are being asked to review the following sections for accuracy:

STUDY DRUG INFORMATION—Please review for accuracy. STUDY DEVICE INFORMATION—Please review for accuracy. RESEARCH ATTRIBUTES—Please review for accuracy. OTHER REVIEW COMMITTEES -- Please review for accuracy.

## **PROJECT INFORMATION**

0 unresolved comment(s)

| Title of Project: (Use the exact title listed in the grant/contract application, if applicable). If your research investigates any aspect of COVID-19, please include "COVID19" at the beginning of your Project Title and Short Title |
|---|
| The Behavioral Effects of Opioids and Alcohol |
| Short Title Description Please use a few key words to easily identify your study - this text will be displayed in the Dashboard listing for your study. Opioids and Alcohol |
| Anticipated Ending Date of Research Project: 6/30/2027 |
| Maximum number of human subjects (or records/specimens to be reviewed) |
| After approval, will the study be open to enrollment of new subjects or new data/specimen collection? ① C Yes 6 No |

Are you requesting that the UK IRB serve as the lead IRB for a multi-site study, **OR** that the UK IRB defer review to another IRB? [Click <u>here</u> for "IRB Reliance" help]

If "Yes," before completing your IRB application, fill out the Reliance Request Form and submit it to irbreliance@uky.edu.

#### PI CONTACT INFORMATION

0 unresolved comment(s)

### Principal Investigator (PI) role for E-IRB access

The PI is the individual holding primary responsibility on the research project with the following permissions on the E-IRB application:

- 1. Read;
- 2. write/edit:
- 3. receive communications; and
- 4. submit to the IRB (IR, CR, MR, Other Review\*).

If research is being submitted to or supported by an extramural funding agency such as NIH, a private foundation or a pharmaceutical/manufacturing company, the PI listed on the grant application or the drug protocol must be listed as PI here.

Please fill in any blank fields with the appropriate contact information (gray shaded fields are not editable). Required fields left blank will be highlighted in pink after you click "Save".

To change home and work addresses, go to myUK and update using the Employee Self Service (ESS) portal. If name has changed, the individual with the name change will need to submit a 'Name Change Form' to the Human Resources Benefits Office for entering into SAP. The new name will need to be associated with the individual's Link Blue ID in SAP before the change is reflected in E-IRB. Contact the HR Benefits Office for additional information.

The Principal Investigator's (PI) contact information is filled in automatically based on who logged in to create the application.

#### If you are not the Principal Investigator, do NOT add yourself as study personnel.

To change the PI contact information on an application in Researcher edit status:

- · click "Change Principal Investigator";
- · search for the PI's name using the search feature;
- click "Select" by the name of the Principal Investigator, then "Save Contact Information".

You will automatically be added as study personnel with editing permissions to continue editing the application.

0

## **Change Principal Investigator:**

| First Name: | Sharon | | Room# &<br>Bldg: | ngliana Avenue |
|---|---|---|---|---|
| Last Name: | Walsh | | Speed<br>Sort#: 1 40508 | 3 |
| Middle Name | L | | | |
| Department: | Behavioral Science - 7H150 | • | Dept Code: 7H15 | 0 |
| Pl's | | | Rank: 🕕 | |
| Employee/Student<br>ID#: | 00058631 | | | Professor |
| PI's Telephone #: | 8592576485 | | Degree: | PhD |
| PI's e-mail<br>address: | sharon.walsh@uky.edu | | PI's FAX<br>Number: | 8592575232 |
| PI is R.N. 🕕 | ⊂ Yes Ģ No | | HSP Trained: | Yes |
| | | | HSP Trained<br>Date: | 1/21/2025 |
| | | | RCR Trained: | Yes |
| Do you, the PI/researcher, have a significant financial interest related to your responsibilities at the University of Kentucky (that requires disclosure per the UK administrative regulation 7:2)? Yes No | | | | |

# RISK LEVEL 0 unresolved comment(s)

Indicate which of the categories listed below accurately describes this protocol

- (Risk Level 1) Not greater than minimal risk
- c (Risk Level 2) Greater than minimal risk, but presenting the prospect of direct benefit to individual subjects
- c (Risk Level 3) Greater than minimal risk, no prospect of direct benefit to individual subjects, but likely to yield generalizable knowledge about the subject's disorder or condition.
- (Risk Level 4) Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of subjects.
- \*"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves from those ordinarily encountered in daily life or during the performance of routine physical or psychological examination or tests.

\*\*\*For Expedited and Exempt Applications, the research activities must be Risk Level 1 (no more than minimal risk to human subjects).\*\*\*

Refer to <u>UK's guidance document</u> on assessing the research risk for additional information.

SUBJECT DEMOGRAPHICS 0 unresolved comment(s)

Age level of human subjects: (i.e., 6 mths.; 2yrs., etc..)  $\boxed{21}$  to  $\boxed{55}$ 

#### **Study Population:**

Describe the characteristics of the subject population, including age range, gender, ethnic background and health status. Identify the criteria for inclusion and exclusion.

Provide the following information:

- A description of the subject selection criteria and rationale for selection in terms of the scientific objectives and proposed study design;
- A compelling rationale for proposed exclusion of any sex/gender or racial/ethnic group;
- Justification for the inclusion of vulnerable groups such as children, prisoners, adults with impaired consent capacity, or others who may be vulnerable to coercion or undue influence.

Please consider this FDA Guidance on Enrollment of Participants from Underrepresented Populations in Clinical Studies



Volunteers will be approximately 72 persons who are screened for the study, with up to 18 (up to 6 pilot participants and up to 12 participants for the fully randomized study) completing the protocol. We anticipate starting recruitment on December 1, 2019, and finishing recruitment by June 30, 2022. Inclusion criteria:

- ages 21-55 years old
- healthy adult male and female participants as determined by physical exam, 12-lead ECG, blood chemistries and routine urinalysis
- recreational (non-medical) opioid use within the past year
- recreational alcohol use within the past year
- must be using an effective form of birth control
- literate and able to provide informed consent
- able and willing to follow the protocol

Exclusion criteria:

- physical dependence on any drug requiring medical management (e.g., opioids, sedatives, alcohol)
- seeking treatment for substance use disorder
- liver function tests exceeding 3x the normal limit
- known hypersensitivity to any of the study drugs
- any psychiatric disorder that would interfere with study participation
- any medical condition that is clinically significant or requires ongoing prescription medication
- acute medical illness unresolved (e.g., infection)
- women who are pregnant or lactating
- current seizure disorder, chronic pain, asthma or other respiratory disorders that may increase risk of respiratory depression
- history of head injury, hypertension, or history of cardiovascular disease or abnormal ECG
- HIV-positive patients if they are symptomatic with AIDS-defining illness (e.g., opportunistic infections, T-cell less than 200/mm3)
- anyone unable to fulfill the protocol requirements based on investigator judgment
- currently under parole or probation with urine testing requirements
- inability to tolerate the pain stimuli during training, reporting no pain/discomfort from cold water test

## Attachments

Indicate the targeted/planned enrollment of the following members of minority groups and their subpopulations. Possible demographic sources: Kentucky State Census, Kentucky Race/Ethnic Table, Kentucky Population Data.

(Please note: The IRB will expect this information to be reported at Continuation Review time for Pre-2019 FDA-regulated Expedited review and Full review applications):

| | | Participant Demo | ographics | |
|---|---|---|---|---|
| | Cisgender Man 🕕 | Cisgender Woman 🕕 | TGNB/TGE 🕕 | Unknown/Not Reported |
| American<br>Indian/Alaskan<br>Native: | | | | |
| Asian: | | | | |
| Black/African<br>American: | 4 | 2 | | |
| Latinx: | 3 | 1 | | |
| Native | | | | |
| Hawaiian/Pacific<br>Islander: | | | | |
| White: | 40 | 20 | | |
| American | | | | |
| Arab/Middle Eastern/North | | | | |
| African: | | | | |
| Indigenous<br>People Around<br>the World: | | | | |

| _ | _ | 4 | _ | • |
|---|---|---|---|----|
| ^ | ` | п | 1 | ıh |

| More than One<br>Race: | 1 | 1 |
|--------------------------|---|---|
| Unknown or Not Reported: | | |

If unknown, please explain why:

Indicate the categories of subjects and controls to be included in the study. You may be required to complete additional forms depending on the subject categories which apply to your research. If the study does not involve direct intervention or direct interaction with subjects, (e.g., record-review research, outcomes registries), do not check populations which the research does not specifically target. For example: a large record review of a diverse population may incidentally include a prisoner or an international citizen, but you should not check those categories if the focus of the study has nothing to do with that status.

-Check All That Apply (at least one item must be selected)-

## ADDITIONAL INFORMATION:

☐ Children (individuals under age

□ Wards of the State (Children)

□ Emancipated Minors

□ Students

□ College of Medicine Students

☐UK Medical Center Residents or

House Officers

□ Impaired Consent Capacity

Adults

☐ Pregnant Women/Neonates/Fetal

Material

□ Prisoners

□ Non-English Speaking (translated long or short form)

□ International Citizens

☐ Military Personnel and/or DoD

Civilian Employees

□ Patients

☐ Appalachian Population

Please visit the <u>IRB Survival Handbook</u> for more information on:

- Children/Emancipated Minors
- Students as Subjects
- Prisoners
- · Impaired Consent Capacity Adults
- Economically or Educationally Disadvantaged Persons

Other Resources:

- UKMC Residents or House Officers [see requirement of GME]
- Non-English Speaking [see also the E-IRB Research Description section on this same topic]
- International Citizens [DoD SOP may apply]
- Military Personnel and/or DoD Civilian Employees

#### Assessment of the potential recruitment of subjects with impaired consent capacity (or likelihood):

Check this box if your study does NOT involve direct intervention or direct interaction with subjects (e.g., record-review research, secondary data analysis). If there is no direct intervention/interaction you will not need to answer the impaired consent capacity questions.

Does this study focus on adult subjects with any conditions that present a high *likelihood* of impaired consent capacity or *fluctuations* in consent capacity? (see examples below)

If Yes and you are not filing for exemption certification, go to "Form T", complete the form, and attach it using the button below.

#### Examples of such conditions include:

- Traumatic brain injury or acquired brain injury
- Severe depressive disorders or Bipolar disorders
- Schizophrenia or other mental disorders that

involve serious cognitive disturbances

- Stroke
- Developmental disabilities
- Degenerative dementias
- CNS cancers and other cancers with possible CNS involvement
- Late stage Parkinson's Disease

- Late stage persistent substance dependence
- Ischemic heart disease
- HIV/AIDS
- COPD
- Renal insufficiency
- Diabetes
- Autoimmune or inflammatory disorders
- Chronic non-malignant pain disorders
- Drug effects
- · Other acute medical crises



#### INFORMED CONSENT/ASSENT PROCESS/WAIVER

0 unresolved comment(s)

For creating your informed consent attachment(s), please download the most up-to-date version listed in "All Templates" under the APPLICATION LINKS menu on the left, and edit to match your research project.

## Additional Resources:

- Informed Consent/Assent Website
- · Waiver of Consent vs. Waiver of Signatures
- Sample Repository/Registry/Bank Consent Template

## Consent/Assent Tips:

- If you have multiple consent documents, be sure to upload each individually (not all in a combined file).
- If another site is serving as the IRB for the project, attach the form as a "Reliance Consent Form" so the document will not receive a UK IRB approval stamp; the reviewing IRB will need to stamp the consent forms.
- Changes to consent documents (e.g., informed consent form, assent form, cover letter, etc...) should be reflected in a 'tracked changes' version and uploaded separately with the Document Type "Highlighted Changes".
- It is very important that only the documents you wish to have approved by the IRB are attached; DELETE OUTDATED FILES -- previously approved versions will still be available in Protocol History.
- Attachments that are assigned a Document Type to which an IRB approval stamp applies will be considered the version(s) to be
  used for enrolling subjects once IRB approval has been issued.
  Document Types that do NOT get an IRB approval stamp are:
  - "Highlighted Changes",
  - "Phone Script", and
  - "Reliance Consent Form",
  - "Sponsor's Sample Consent Form".

#### How to Get the Section Check Mark

- 1. You must:
  - a) provide a response in the text box below describing how investigators will obtain consent/assent, and
  - b) check the box for at least one of the consent items and/or check mark one of the waivers
- 2. If applicable attach each corresponding document(s) as a read-only PDF.
- 3. If you no longer need a consent document approved (e.g., closed to enrollment), or, the consent document submitted does not need a stamp for enrolling subjects (e.g., umbrella study, or sub-study), only select "Stamped Consent Doc(s) Not Needed".
- 4. After making your selection(s) be sure to scroll to the bottom of this section and SAVE your work!



#### -Check All That Apply-

- □ Informed Consent Form (and/or Parental Permission Form and/or translated short form)
- ☐ Assent Form
- □ Cover Letter (for survey/questionnaire research)
- ☐ Phone Script
- □Informed Consent/HIPAA Combined Form
- □ Debriefing and/or Permission to Use Data Form
- □ Reliance Consent Form
- □ Sponsor's sample consent form for Dept. of Health and Human Services (DHHS)-approved protocol



## **Informed Consent Process:**

Using active voice, in the text box below, describe how investigators will obtain consent/assent. Include:

- the circumstances under which consent will be sought and obtained
- · the timing of the consent process (including any waiting period between providing information and obtaining consent)

- · who will seek consent
- how you will minimize the possibility of coercion or undue influence
- the method used for documenting consent
- if applicable, who is authorized to provide permission or consent on behalf of the subject
- if applicable, specific instruments or techniques to assess and confirm potential subjects' understanding of the information

Will electronic consent form/process be utilized on-site or remotely for this study?

∩ Yes ∩ No

If yes, in addition to addressing the above bullet points, describe the e-consent method and platform, including any hyperlinks, videos, or enhancements used to convey information, if applicable. Attach a representation of the e-consent with signature fields. For guidance, see the ORI <u>E-Consent web page</u>.

Note: all individuals authorized to obtain informed consent should be designated as such in the E-IRB "Study Personnel" section of this application.

Special considerations may include:

- Obtaining consent/assent for special populations such as children, prisoners, or people with impaired decisional capacity
- Research Involving Emancipated Individuals
   If you plan to enroll some or all prospective subjects as emancipated, consult with UK legal counsel prior to submitting this application to the IRB. Include research legal counsel's recommendations in the "Additional Information" section as a separate document.
- Research Involving Non-English Speaking Subjects
   For information on inclusion of non-English speaking subjects, or subjects from a foreign culture, see IRB Application Instructions for Recruiting Non-English Speaking Participants or Participants from a Foreign Culture.
- Research Repositories

If the purpose of this submission is to establish a research repository describe the informed consent process. For guidance regarding consent issues, process approaches, and sample language see the <a href="Sample Repository/Registry/Bank Consent Template">Sample Repository/Registry/Bank Consent Template</a>.

Prior to obtaining informed consent, each potential subject must have an expired breath alcohol content (BAC) of 0.00 and not appeared intoxicated (nodding, appearing sedated). Sharon L. Walsh, Ph.D. or her designated staff will obtain consent for this project. There are two consent forms for this project: a screening consent and the main study consent. Designated staff may conduct and sign the informed screening consent with the volunteer. However, the volunteer will meet with an investigator or senior staff member prior to admission to review all experimental procedures and allow the volunteer ample time to ask questions regarding the protocol before signing the study consent form. There is no time limit on this process. The investigator will inform the volunteer that this is not a treatment program and signing the consent form does not obligate them to participate. Each subject will receive a copy of his/her informed consent document.

Participants may also be consented via Zoom. All consenting procedures will be identical to an in-person consent, except the PI will be present via Zoom (instead of the same room). The participant will be screened by in-person research staff (e.g., participants provided photo ID, negative breathalyzer samples and protocol-appropriate urine samples; staff confirmed participants were not intoxicated). Research staff will provide the a copy of the hardcopy (paper) consent form to the participant, which will be verified on camera by the PI. This process allows for a thorough discussion and exchange of information with the participant, a method to ensure the participant's identity, and documentation of the consent itself.

Subjects may ask study personnel questions about the study procedures or make complaints at any time. All staff will be aware to contact the Principal Investigator, Sharon Walsh, Ph.D., about any subject concern or complaint as it arises. Phone numbers for the PI and medically responsible investigator as well as the Office of Research Integrity, are included in the consent form. It is expected that providing a phone number and contact information for the PI may offer a safe, confidential and reliable channel for participants to express problems, concerns or questions and obtain study information.

□ Request for Waiver of Informed Consent Process

If you are requesting IRB approval to waive the requirement for the informed consent process, or to alter some or all of the elements of informed consent, complete, Section 1 and Section 2 below.

Note: The IRB does not approve waiver or alteration of the consent process for greater than minimal risk research, except for planned emergency/acute care research as provided under FDA regulations. Contact ORI for regulations that apply to single emergency use waiver or acute care research waiver (859-257-9428).

## **SECTION 1.**

Check the appropriate item:

■ I am requesting a waiver of the requirement for the informed consent process.

■I am requesting an alteration of the informed consent process.

If you checked the box for this item, describe which elements of consent will be altered and/or omitted, and justify the

alteration.

## **SECTION 2.**

Explain how each condition applies to your research.

- a) The research involves no more than minimal risk to the subject.
- b) The rights and welfare of subjects will not be adversely affected.
- c) The research could not practicably be carried out without the requested waiver or alteration.
- d) Whenever possible, the subjects or legally authorized representatives will be provided with additional pertinent information after they have participated in the study.
- e) If the research involves using or accessing identifiable private information or identifiable biospecimens, the research could not practicably be carried out without using such information or biospecimens in an identifiable format.
  - Private information/specimens are "identifiable" if the investigator may ascertain the identity of the subject or if identifiers
    are associated with the information (e.g., medical records). This could be any of the <u>18 HIPAA identifiers</u> including <u>dates</u>
    of service.
  - If not using identifiable private information or identifiable biospecimens, insert N/A below.

If you are requesting IRB approval to waive the requirement for signatures on informed consent forms, **your research** activities must fit into one of three regulatory options:

- 1. The only record linking the participant and the research would be the consent document, and the principal risk would be potential harm resulting from a breach of confidentiality (e.g., a study that involves participants who use illegal drugs).
- 2. The research presents no more than minimal risk to the participant and involves no procedures for which written consent is normally required outside of the research context (e.g., a cover letter on a survey, or a phone script).
- 3. The participant (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm, the research presents no more than minimal risk to the subject, and there is an appropriate alternative mechanism for documenting that informed consent was obtained.

Select the option below that best fits your study.

If the IRB approves a waiver of signatures, participants must still be provided oral or written information about the study. To ensure you include required elements in your consent document, use the **Cover Letter Template** as a guide. There is an <u>English</u> and a <u>Spanish</u> version.



## Option 1

## Describe how your study meets these criteria:

- a) The only record linking the participant and the research would be the consent document:
- b) The principal risk would be potential harm resulting from a breach of confidentiality (i.e., a study that involves subjects who use illegal drugs).

Under this option, each participant (or legally authorized representative) must be asked whether (s)he wants to sign a consent document; if the participant agrees to sign a consent document, only an IRB approved version should be used.

## COption 2

## Describe how your study meets these criteria:

- a) The research presents no more than minimal risk to the participant:
- b) Involves no procedures for which written consent is normally required outside of the research context (i.e. a cover letter on a survey, or a phone script):

## © Option 3

#### Describe how your study meets these criteria:

- a) The subject (or legally authorized representative) is a member of a distinct cultural group or community in which signing forms is not the norm.
- b) The research presents no more than minimal risk to the subject.
- c) There is an appropriate alternative mechanism for documenting that informed consent was obtained.

#### STUDY PERSONNEL 0 unresolved comment(s)

Do you have study personnel who will be assisting with the research?

After selecting 'Yes' or 'No' you must click the 'Save Study Personnel Information' button.

c Yes c No

#### Manage Study Personnel

Identify other study personnel assisting in research project:

- The individual listed as PI in the 'PI Contact Information' section should NOT be added to this section.
- If the research is required for a University of Kentucky academic program, the faculty advisor is also considered study personnel and should be listed below. \*\*\*Residents and students who are PI's are encouraged to designate the faculty advisor or at least one other individual as a contact with an editor role (DP).\*\*\*
- Role: DP = Editor (individual can view, navigate, and edit the application for any review phase (IR, CR/FR, MR) or 'Other Review", and submit Other Reviews on behalf of the Pl.)
- Role: SP = Reader (individual can view and navigate through the currently approved application only.)

To add an individual via the below feature:

- · Search for personnel;
- Click "select" by the listing for the person you want to add;
- For each person, specify responsibility in the project, whether authorized to obtain informed consent, AND denote who should receive E-IRB notifications (contact status).

NOTE: Study personnel must complete human subject protection (HSP) and Responsible Conduct of Research (RCR) training before implementing any research procedures. For information about training requirements for study personnel, visit UK's <a href="https://example.com/HSP FAQ page">HSP FAQ page</a>, the <a href="https://example.com/RCR HSP training cher than that acquired through UK CITI, you may submit it to ORI (<a href="https://example.com/HSPTrainingSupport@uky.edu">HSPTrainingSupport@uky.edu</a>) for credit.

#### Study personnel assisting in research project: 0

| Last Name | First Name | Responsibility In<br>Project | Role | A<br>C | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | Last<br>Updated | SFI | Active |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Andrews | Lelia | Data Collection | SP | Υ | N | | Р | Υ | 01/20/2023 | Υ | N | 01/19/2023 | N | Υ |
| Babalonis | Shanna | Co-Investigator | DP | Υ | Υ | PhD | Р | Υ | 06/04/2024 | Υ | N | 11/11/2019 | Ν | Υ |
| Canedo | Anabel | Data Collection | SP | Υ | N | | S | Υ | 07/13/2025 | Υ | N | 07/14/2025 | N | Υ |
| Christian | Eli | Data Collection | SP | Υ | N | | Р | Υ | 04/17/2024 | Υ | N | 04/18/2024 | N | Υ |
| Dowden-<br>Kruger | Melinda | Project<br>Assistance/Support | DP | N | Υ | | Р | Υ | 09/27/2024 | Υ | N | 11/06/2019 | N | Υ |
| Fanucchi | Laura | Medical Supervisor | SP | Υ | N | MD,<br>MPH | Р | Υ | 01/17/2025 | Υ | N | 11/11/2019 | N | Υ |
| Fuller | Grayson | Data Collection | SP | Υ | N | | Р | Υ | 03/15/2023 | Υ | N | 03/16/2023 | N | Υ |
| Hash | Matthew | Project<br>Assistance/Support | SP | N | N | | Р | Υ | 01/26/2024 | Υ | N | 03/13/2020 | N | Υ |
| Hunt | Cassandra | Data Collection | SP | N | N | | Р | Υ | 02/12/2024 | Υ | N | 03/13/2020 | N | Υ |
| Lofwall | Michelle | Medical Supervisor | SP | Υ | N | MD | Р | Υ | 06/29/2023 | Υ | N | 11/11/2019 | N | Υ |
| Murphy | John | Consultant/Advisor | SP | N | N | | Р | Υ | 08/12/2025 | Υ | N | 03/13/2020 | N | Υ |
| Nuzzo | Paul | Data<br>Analysis/Processing | SP | Υ | N | MA | Р | Υ | 01/30/2023 | Υ | N | 11/11/2019 | N | Υ |
| Perpar | Justin | Data Collection | SP | Υ | N | | Р | Υ | 10/26/2022 | Υ | N | 10/26/2022 | Ν | Υ |
| Randolph | Carly | Data Collection | SP | Υ | N | | S | Υ | 06/14/2024 | Υ | N | 06/17/2024 | N | Υ |
| Stafford | Maribeth | Data Collection | SP | Υ | N | | S | Υ | 07/19/2023 | Υ | N | 05/28/2024 | Ν | Υ |
| VanMeter | Connor | Data Collection | SP | Υ | N | | Р | Υ | 04/14/2025 | Υ | N | 10/28/2021 | N | Υ |
| Vessels | Victoria | Data Collection | SP | Υ | N | | Р | Υ | 05/02/2025 | Υ | N | 11/11/2019 | Ν | Υ |
| AbouAhmed | Amira | Data Collection | SP | Ν | N | | Р | N | 10/22/2019 | | Υ | 04/29/2022 | Ν | Ν |
| Adams | Christian | Medical Supervisor | SP | N | N | MD | Р | Υ | 12/21/2022 | Υ | Υ | 01/27/2025 | Ν | Υ |
| Adams | Elizabeth | Data Collection | SP | Ν | N | RN | Р | N | 10/22/2020 | | Υ | 04/29/2022 | Ν | N |
| Ali | Nur-Ur-<br>Sahar | Data Collection | SP | Υ | N | | Р | N | 08/06/2020 | | Υ | 08/04/2021 | N | N |
| Allen | Nicola | Data Collection | SP | Ν | N | RN | Р | N | 10/29/2020 | Υ | Υ | 02/03/2023 | N | N |
| Allen | Remi | Data Collection | SP | Υ | N | | S | N | 07/17/2019 | | Υ | 06/24/2020 | N | Υ |
| Allen | Timothy | Medical Supervisor | SP | N | N | MD | Р | Υ | 12/04/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| Anderson | Danielle | Medical Supervisor | SP | N | N | MD | Р | Υ | 05/31/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| Antel | Mallory | Data Collection | SP | Υ | N | | Р | N | 07/22/2019 | Υ | Υ | 10/14/2020 | N | N |
| Atwater | Chelsea | Medical Supervisor | SP | N | N | MD | Р | Υ | 10/25/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| Bailey | Rebecca | Data Collection | SP | Ν | N | RN | Р | Υ | 09/08/2022 | Υ | Υ | 01/21/2025 | N | Υ |
| Bailey-Offill | Emilee | Medical Supervisor | SP | N | N | MD | S | N | 08/29/2017 | | Υ | 10/14/2020 | N | N |
| Batsel-<br>Thomas | Sandra | Medical Supervisor | SP | N | N | MD | Р | Υ | 06/03/2024 | Υ | Υ | 01/27/2025 | N | Υ |

| Desirable Amantan Data Collection SP N N N N N N N N N | | | | | | | | | | | | | | JJ 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Berlein | Last Name | First Name | | Role | | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | | SFI | Active |
| Belacht Black | Binkley | Amanda | Data Collection | SP | Υ | N | RN | Р | N | 04/10/2018 | | Υ | 03/13/2020 | N | N |
| Browne | Bradley | Robin | Data Collection | SP | N | N | RN | Р | N | 05/24/2019 | | Υ | 09/22/2022 | N | N |
| Brown | Britch | Stevie | Co-Investigator | DP | Υ | Υ | | Р | N | 07/29/2022 | Υ | Υ | 07/28/2023 | N | N |
| Brown | Broome | Bibi | Data Collection | SP | N | N | | Р | Υ | 03/21/2023 | Υ | Υ | 04/29/2022 | N | Υ |
| Brushing | Brown | Paul | Data Collection | SP | N | N | | Р | Υ | 09/08/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Buckler Regan Data Collection SP N N RN P Y O4/16/20124 Y Y O1/23/2025 N Y Casy | Brown | Vickie | Data Collection | SP | N | N | RN | Р | N | 02/14/2020 | Υ | Υ | 02/28/2023 | N | Υ |
| Campy Contest | Browning | Christopher | Data Collection | SP | N | N | | Р | Υ | 09/18/2023 | Υ | Υ | 10/18/2022 | N | Υ |
| Camper Zemith Data Collection SP N N RN P Y 02/18/2023 Y Y 01/23/2025 N N Champal Load Data Collection SP N N RN P Y 02/17/2026 Y Y 01/23/2025 N Y Champal Load Data Collection SP N N RN P Y 02/17/2023 Y Y 01/23/2025 N Y Champal Load Collection SP N N RN P Y 03/26/2023 Y Y 01/23/2025 N Y Clark Kate Data Collection SP N N RN P Y 03/26/2023 Y Y 01/23/2025 N Y Clark Kate Data Collection SP N N RN P Y 03/26/2024 Y Y 07/28/2023 N N Cobb Sasam Data Collection SP N N RN P Y 03/26/2024 Y Y 01/23/2025 N Y Cocle Mark Data Collection SP N N MD P Y 03/26/2024 Y Y 01/27/2025 N Y Cocle Mark Data Collection SP N N RN P N 03/37/2022 Y Y 01/27/2025 N Y Davino Arabew Data Collection SP N N RN P N 03/37/2022 Y Y 06/18/2025 N Y Davino Arabew Data Collection SP N N RN P N 03/37/2022 Y Y 06/18/2025 N Y Davino Arabew Data Collection SP N N RN P N 03/37/2022 Y Y 06/18/2023 N N Ethir Kathritim Data Collection SP N N RN P N 03/37/2022 Y Y 01/18/2022 N Y Ethir Kathritim Data Collection SP N N RN P Y 05/17/2023 Y Y 07/26/2023 N N Ethir Kathritim Data Collection SP N N RN P Y 05/17/2023 Y Y 02/26/2023 N N Ethir Carle Data Collection SP N N RN P Y 05/17/2023 Y Y 02/26/2023 N N Ethir Carle Data Collection SP N N RN P Y 05/17/2023 Y Y 07/26/2025 N Y Ethir Data Collection SP N N RN P Y 05/17/2023 Y Y 06/26/2022 N Y Ethir Data Collection SP N N RN P Y 05/17/2023 Y Y 06/26/2022 N Y Ethir Data Collection SP N N RN P Y 05/17/2023 Y Y 01/23/2025 N Y Ethir Data Co | Buckler | Regan | Data Collection | SP | N | N | RN | Р | Υ | 04/16/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Chamble Lisa | Cady | Corissa | Data Collection | SP | N | N | | Р | Υ | 06/05/2023 | Υ | Υ | 01/23/2025 | N | N |
| Chiang Loi Data Collection SP Y N P Y 08/08/2023 Y Y 01/21/2025 N N Chiang Ebabeth Data Collection SP N N P Y 09/22/2023 Y Y 01/23/2025 N Y Clark Clark Katle Data Collection SP N N RN P Y 09/22/2023 Y Y 01/23/2025 N Y Clark Cl | Camper | Zenith | Data Collection | SP | N | N | RN | Р | Υ | 02/08/2023 | Υ | Υ | 01/23/2025 | N | N |
| Chillian Elizabelin Data Collection SP N N P Y 09/28/2023 Y Y 01/23/2025 N Y Clark Katile Data Collection SP Y N P Y 01/10/2022 Y Y 07/28/2023 N N Cobb Susan Data Collection SP N N FN P Y 01/30/2022 Y Y 07/28/2023 N N Cobb Susan Data Collection SP N N FN P Y 01/30/2024 Y Y 07/28/2023 N N Code Manco Data Collection SP N N MD P Y 12/29/2023 Y Y 01/27/2025 N Y Thirting | Chamblin | Lisa | Data Collection | SP | Ν | N | RN | Р | Υ | 07/17/2025 | Υ | Υ | 01/23/2025 | Ν | Υ |
| Clark Kate Data Collection SP Y N P Y 10/10/2022 Y Y 07/28/2023 N N Cobb Susan Data Collection SP N N RN P Y 0.3/30/2024 Y Y 01/23/2025 N Y Code Merion Data Collection SP Y N P N 11/30/2016 Y 11/11/2019 N Y Code Y Y 0.1/23/2025 N Y Y Code Y Y Toda Y Y Toda Y Y Toda Y Y Toda Y Y Toda Y Y Toda Y Y Y Y Y Y Y Y Y | Chang | Loui | Data Collection | SP | Υ | N | | | Υ | 06/05/2023 | Υ | Υ | 01/21/2025 | N | N |
| Cobb Susan Data Collection SP N N FN P Y 03/30/2024 Y Y 01/23/2025 N Y Code Marton Data Collection SP Y N P N 11/03/2016 Y 11/13/2019 N N N N P N 11/03/2016 Y 11/13/2019 N N N N P N 11/03/2016 Y 11/13/2019 N N N N N P N 11/03/2021 Y Y 01/23/2025 N Y N N N P N 08/31/2022 Y Y 01/23/2025 N Y N N N P N 08/31/2022 Y Y 01/23/2025 N Y N N N P N 08/31/2022 Y Y 08/28/2023 N N N N N P N 08/31/2022 Y Y 08/28/2023 N N N N N N P N 05/30/2019 Y 11/04/2021 N N N N N N N N N | Chilton | Elizabeth | Data Collection | SP | N | N | | Р | Υ | 09/28/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Coe | Clark | Katie | Data Collection | SP | Υ | N | | Р | Υ | 10/10/2022 | Υ | Υ | 07/28/2023 | N | N |
| Cooley | Cobb | Susan | Data Collection | SP | N | N | RN | Р | Υ | 03/30/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Davis Miranda Data Collection SP Y N FN P N 08/31/2022 Y Y 06/18/2025 N Y | Coe | Marion | Data Collection | SP | Υ | N | | Р | N | 11/03/2016 | | Υ | 11/11/2019 | N | N |
| Devine | Cooley | Andrew | Medical Supervisor | SP | N | N | MD | Р | Υ | 12/29/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| Dugan Joseph Data Collection SP N N RN P N 05/30/2019 Y 10/04/2021 N N Edmiston Emily Data Collection SP Y N MPH P N 10/16/2017 Y 11/11/2018 N N Elder Katherine Data Collection SP N N RN P Y 05/31/2024 Y Y 10/18/2022 N Y Erp Joyce Data Collection SP N N RN P Y 05/31/2024 Y Y 01/23/2025 N Y Y Y Y Y Y Y Y Y | Davis | Miranda | Data Collection | SP | Υ | N | RN | Р | N | 08/31/2022 | Υ | Υ | 06/18/2025 | N | Υ |
| Edmiston Emily Data Collection SP Y N MPH P N 10/16/2017 Y 11/11/2019 N N Elder Katherine Data Collection SP N N S Y 09/24/2024 Y Y 10/18/2022 N Y 10/18/2023 N N P N N RN P Y 05/21/2023 Y Y 02/28/2023 N N P N RN P Y 05/21/2023 Y Y 02/28/2023 N N P N RN P Y 05/21/2023 N Y 10/18/2022 N Y 10/18/2023 N N P N N RN P Y 05/24/2024 Y Y 01/28/2023 N N P N RN P N 08/08/2022 Y Y 01/28/2023 N N P N RN P N 08/08/2022 Y Y 01/28/2023 N N P N RN P N 08/08/2022 Y Y 01/28/2023 N N P N RN P N 08/08/2022 Y Y 01/28/2023 N N P N RN P N 08/08/2024 Y Y 01/28/2022 N Y N N RN P N N RN P N 08/08/2024 Y Y 01/28/2022 N Y 01/28/2022 N Y N N RN P N 08/08/2024 Y Y 01/28/2022 N Y 0 | Devine | Amber | Data Collection | SP | N | N | | Р | N | 11/23/2021 | Υ | Υ | 06/28/2023 | N | N |
| Elder Katherine Dafa Collection SP N N S Y 09/24/2024 Y Y 10/18/2022 N Y | Dugan | Joseph | Data Collection | SP | N | N | RN | Р | N | 05/30/2019 | | Υ | 10/04/2021 | N | N |
| Erp Joyce Data Collection SP N N RN P Y 05/31/2024 Y Y 01/23/2025 N Y Evans Rachel Data Collection SP N N RN P Y 05/21/2023 Y Y 02/21/2024 N N Famel Carla Data Collection SP N N RN P Y 01/17/2023 Y Y 02/28/2023 N N Fayne Kristen Data Collection SP N RN P Y 01/17/2023 Y Y 04/24/2022 N Y Finch Megan Data Collection SP N N RN P Y 05/24/2024 Y Y 01/23/2025 N Y Finch Megan Data Collection SP N N RN P Y 02/22/2023 Y 06/28/2023 N N < | Edmiston | Emily | Data Collection | SP | Υ | N | MPH | Р | N | 10/16/2017 | | Υ | 11/11/2019 | N | N |
| Evans Rachel Data Collection SP N RN P Y 05/21/2023 Y Q:/01/2024 N N Fancher Joshua Data Collection SP Y N P Y 01/17/2023 Y Y 02/28/2023 N N Farrell Carla Data Collection SP N N RN P Y 10/11/2024 Y Q:/04/2022 N Y Fayne Kristan Data Collection SP N N RN P Y 05/24/2024 Y Q:/01/23/2025 N Y Finch Megan Data Collection SP N N RN P Y 02/02/2023 Y Q:/01/23/2025 N Y Fortz Denise Project SP N N RN P Y 02/02/2023 Y Q:/01/23/2025 N Y Gamble Bethanie Data Collection | Elder | Katherine | Data Collection | SP | N | N | | S | Υ | 09/24/2024 | Υ | Υ | 10/18/2022 | N | Υ |
| Fancher Joshua Data Collection SP Y N P Y 01/17/2023 Y Y 02/28/2023 N N Farrell Carla Data Collection SP N N RIN P Y 10/11/2024 Y Q 04/04/2022 N Y Fayne Kristen Data Collection SP N N RIN P Y 05/24/2024 Y 04/04/2022 N Y Finch Megan Data Collection SP N N RN P Y 05/24/2024 Y 06/28/2023 N N Foritz Denise Project Project SP N N RN P Y 02/02/2023 Y 06/18/2023 N Y Foritz Denise Project SP N N RN P Y 02/02/2023 Y 05/11/2023 N 0 05/11/2023 Y | Erp | Joyce | Data Collection | SP | N | N | RN | Р | Υ | 05/31/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Farrell Carla Data Collection SP N N RN P Y 10/11/2024 Y 04/04/2022 N Y Fayne Kristen Data Collection SP N N RN P Y 05/24/2024 Y 01/23/2025 N Y Finch Megan Data Collection SP N N P N 08/08/2022 Y 06/28/2023 N N Foltz Denise Project<br>Assistance/Support SP N N RN P Y 02/20/2023 Y 05/17/2023 N Y Forenback Denise Project<br>Assistance/Support SP N RN P Y 12/20/2023 Y 05/17/2023 N Y Gamble Bethanie Data Collection SP N RN P N 09/07/2021 Y 01/23/2025 N Y Garton Jackson Data Collection S | Evans | Rachel | Data Collection | SP | N | N | RN | Р | Υ | 05/21/2023 | Υ | Υ | 02/01/2024 | N | N |
| Fayne Kristen Data Collection SP N RN P Y 05/24/2024 Y Y 01/23/2025 N Y Finch Megan Data Collection SP N N P N 08/08/2022 Y Y 06/28/2023 N N Foltz Denise Project<br>Assistance/Support SP Y N P Y 02/02/2023 Y Y 05/17/2023 N Y Forenback Denece Data Collection SP N R P Y 12/07/2023 Y Y 01/23/2025 N Y Gamble Data Collection SP N R N R P Y 10/03/2022 Y 07/08/2024 N N Garden Jackson Data Collection SP N R N P N 09/24/2021 Y Y 01/23/2025 N Y Garden Jack | Fancher | Joshua | Data Collection | SP | Υ | N | | Р | Υ | 01/17/2023 | Υ | Υ | 02/28/2023 | N | N |
| Finch Megan Data Collection SP N N P N 08/08/2022 Y Y 06/28/2023 N N Foltz Denise Project<br>Assistance/Support SP Y N P Y 02/02/2023 Y Y 05/17/2023 N Y Forenback Denece Data Collection SP N N RN P Y 12/07/2023 Y Y 01/23/2025 N Y Gamble Bethanie Data Collection SP N N RN P Y 10/03/2022 Y Y 07/09/2024 N N Garnett Kimberty Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Garton Jackson Data Collection SP N N RN P N 09/07/2021 Y 01/29/2022 N Y <td>Farrell</td> <td>Carla</td> <td>Data Collection</td> <td>SP</td> <td>N</td> <td>N</td> <td>RN</td> <td>Р</td> <td>Υ</td> <td>10/11/2024</td> <td>Υ</td> <td>Υ</td> <td>04/04/2022</td> <td>N</td> <td>Υ</td> | Farrell | Carla | Data Collection | SP | N | N | RN | Р | Υ | 10/11/2024 | Υ | Υ | 04/04/2022 | N | Υ |
| Foltz Denise Project Assistance/Support SP Y N P P Y 02/02/2023 Y Y 05/17/2023 N Y Forenback Denece Data Collection SP N N RN P Y 12/07/2023 Y Y 01/23/2025 N Y Gamble Bethanie Data Collection SP N N RN P Y 10/03/2022 Y Y 07/08/2024 N N RAN P N 09/07/2021 Y Y 07/08/2024 N N Garnett Kimberly Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Garton Jackson Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Garton Jackson Data Collection SP N N RN P N 09/24/2021 Y Y 01/23/2025 N Y Gayhart Sarah Data Collection SP N N RN P Y 09/21/2023 Y Y 01/23/2025 N Y Gevedon Teresa Medical Supervisor SP N N MD P N 06/01/2022 Y Y 05/11/2021 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P N 09/04/2021 Y Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP N N RN P N 05/08/2017 Y 11/13/2019 N N GONZález-Lozano Evelyn Data Collection SP N N RN P N 05/08/2017 Y 11/13/2019 N N Harmi Anna Data Collection SP N N RN P N 09/21/2024 Y Y 10/09/2024 N Y Harmi Shontel Data Collection SP N N RN P N 09/21/2024 Y Y 10/09/2024 N Y Harmi Shontel Data Collection SP N N RN P N 09/21/2024 Y Y 10/09/2024 N Y Harmi Shontel Data Collection SP N N RN P N 09/21/2024 Y Y 10/09/2024 N Y Harmi Shontel Data Collection SP N N MD P Y 09/21/2024 Y Y 01/27/2025 N Y 14/200 Medical Supervisor SP N N MD P Y 09/21/2024 Y Y 01/27/2025 N Y 14/200 Medical Supervisor SP N N MD P Y 09/21/2024 Y Y 01/27/2025 N Y 14/200 Medical Supervisor SP N N MD P Y 09/21/2024 Y Y 01/27/2025 N Y 14/200 Medical Supervisor SP N N MD P Y 09/21/2024 Y Y 01/27/2025 N Y 01/27/2025 | Fayne | Kristen | Data Collection | SP | N | N | RN | Р | Υ | 05/24/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Folize | Finch | Megan | | SP | N | N | | Р | N | 08/08/2022 | Υ | Υ | 06/28/2023 | N | N |
| Gamble Bethanie Data Collection SP N RN P Y 10/03/2022 Y Y 07/08/2024 N N Garnett Kimberly Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Garnett Kimberly Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Gardon Jackson Data Collection SP N N RN P N 09/07/2021 Y Y 01/23/2025 N Y Gayhart Sarah Data Collection SP N N MD P Y 09/21/2023 Y Y 01/123/2025 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y 01/23/2025 N Y | Foltz | Denise | • | SP | Υ | N | | Р | Υ | 02/02/2023 | Υ | Υ | 05/17/2023 | N | Υ |
| Garnett Kimberly Data Collection SP N N RN P N 09/07/2021 Y Y 04/29/2022 N Y Garton Jackson Data Collection SP Y N P N 09/24/2021 Y Y 10/28/2021 N Y Garyhart Sarah Data Collection SP N N RN P Y 09/21/2023 Y Y 01/23/2025 N Y Gevedon Teresa Medical Supervisor SP N N MD P N 06/01/2022 Y Y 05/11/2021 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 01/23/2022 N Y< | Forenback | Denece | Data Collection | SP | Ν | N | RN | Р | Υ | 12/07/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Garton Jackson Data Collection SP Y N P N 09/24/2021 Y Y 10/28/2021 N Y Gayhart Sarah Data Collection SP N N RN P Y 09/21/2023 Y Y 01/23/2025 N Y Gevedon Teresa Medical Supervisor SP N N MD P N 06/01/2022 Y Y 05/11/2021 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Gollamudi Anusha Data Collection SP N N P N 05/08/2017 Y 11/13/2019 N N <t< td=""><td>Gamble</td><td>Bethanie</td><td>Data Collection</td><td>SP</td><td>Ν</td><td>N</td><td>RN</td><td>Р</td><td>Υ</td><td>10/03/2022</td><td>Υ</td><td>Υ</td><td>07/08/2024</td><td>N</td><td>N</td></t<> | Gamble | Bethanie | Data Collection | SP | Ν | N | RN | Р | Υ | 10/03/2022 | Υ | Υ | 07/08/2024 | N | N |
| Gayhart Sarah Data Collection SP N RN P Y 09/21/2023 Y Y 01/23/2025 N Y Gevedon Teresa Medical Supervisor SP N N MD P N 06/01/2022 Y Y 05/11/2021 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P Y 10/02/2024 Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP N N P N 05/08/2017 Y 11/13/2019 N N Gonzalez-<br>Lozano< | Garnett | Kimberly | Data Collection | SP | N | N | RN | Р | N | 09/07/2021 | Υ | Υ | 04/29/2022 | N | Υ |
| Gevedon Teresa Medical Supervisor SP N N MD P N 06/01/2022 Y Y 05/11/2021 N Y Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P Y 10/02/2024 Y Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP N N P N 05/08/2017 Y 11/13/2019 N N Gorzalez-Lozano Evelyn Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N | Garton | Jackson | Data Collection | SP | Υ | N | | Р | N | 09/24/2021 | Υ | Υ | 10/28/2021 | N | Υ |
| Gibson Pamela Data Collection SP N N RN P Y 07/27/2023 Y Y 01/23/2025 N Y Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P Y 10/02/2024 Y Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP Y N P N 05/08/2017 Y 11/13/2019 N N Gonzalez-Lozano Evelyn Data Collection SP Y N P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N | Gayhart | Sarah | Data Collection | SP | N | N | RN | Р | Υ | 09/21/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Gifford Mariah Data Collection SP N N RN P N 09/04/2021 Y Y 04/29/2022 N Y Golenbiewski Nicole Data Collection SP N N RN P Y 10/02/2024 Y Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP Y N P N 05/08/2017 Y 11/13/2019 N N Gonzalez-Lozano Evelyn Data Collection SP Y N P P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Hatris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP N N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Gevedon | Teresa | Medical Supervisor | SP | N | N | MD | Р | N | 06/01/2022 | Υ | Υ | 05/11/2021 | N | Υ |
| Golenbiewski Nicole Data Collection SP N N RN P Y 10/02/2024 Y Y 01/23/2025 N Y Gollamudi Anusha Data Collection SP Y N P N 05/08/2017 Y 11/13/2019 N N Gonzalez-Lozano Evelyn Data Collection SP Y N P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Harris Shontel Data Collection SP N N MD P Y 09/21/2024 Y Y 10/09/2024 N Y | Gibson | Pamela | Data Collection | SP | Ν | N | RN | Р | Υ | 07/27/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Gollamudi Anusha Data Collection SP Y N P N 05/08/2017 Y 11/13/2019 N N Gonzalez-Lozano Evelyn Data Collection SP Y N P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Harris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP N N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne | Gifford | Mariah | Data Collection | SP | Ν | N | RN | Р | N | 09/04/2021 | Υ | Υ | 04/29/2022 | N | Υ |
| Gonzalez-Lozano Evelyn Data Collection SP Y N P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Harris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP Y N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y <td>Golenbiewski</td> <td>Nicole</td> <td>Data Collection</td> <td>SP</td> <td>N</td> <td>N</td> <td>RN</td> <td>Р</td> <td>Υ</td> <td>10/02/2024</td> <td>Υ</td> <td>Υ</td> <td>01/23/2025</td> <td>N</td> <td>Υ</td> | Golenbiewski | Nicole | Data Collection | SP | N | N | RN | Р | Υ | 10/02/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Lozano Evelyn Data Collection SP Y N P Y 07/09/2024 Y Y 10/09/2024 N Y Hamilton Rebekah Data Collection SP N N RN P N 10/31/2020 Y 06/14/2022 N N Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Harris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP Y N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y <tr< td=""><td>Gollamudi</td><td>Anusha</td><td>Data Collection</td><td>SP</td><td>Υ</td><td>N</td><td></td><td>Р</td><td>N</td><td>05/08/2017</td><td></td><td>Υ</td><td>11/13/2019</td><td>N</td><td>N</td></tr<> | Gollamudi | Anusha | Data Collection | SP | Υ | N | | Р | N | 05/08/2017 | | Υ | 11/13/2019 | N | N |
| Hamm Anna Data Collection SP N N CNA P Y 03/29/2023 Y Y 10/09/2024 N Y Harris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP Y N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | | Evelyn | Data Collection | SP | Υ | N | | Р | Υ | 07/09/2024 | Υ | Υ | 10/09/2024 | N | Υ |
| Harris Shontel Data Collection SP N N P Y 09/21/2024 Y Y 10/09/2024 N Y Hatton Kevin Medical Supervisor SP Y N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Hamilton | Rebekah | Data Collection | SP | N | N | RN | Р | N | 10/31/2020 | | Υ | 06/14/2022 | N | N |
| Hatton Kevin Medical Supervisor SP Y N MD P Y 08/18/2024 Y Y 01/27/2025 N Y Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Hamm | Anna | Data Collection | SP | N | N | CNA | Р | Υ | 03/29/2023 | Υ | Υ | 10/09/2024 | N | Υ |
| Hawthorne James Medical Supervisor SP N N MD P Y 05/09/2023 Y Y 01/27/2025 N Y Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Harris | Shontel | Data Collection | SP | N | N | | Р | Υ | 09/21/2024 | Υ | Υ | 10/09/2024 | N | Υ |
| Hays Lon Medical Supervisor SP N N MD P Y 11/08/2023 Y Y 01/27/2025 N Y Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Hatton | Kevin | Medical Supervisor | SP | Υ | N | MD | Р | Υ | 08/18/2024 | Υ | Υ | 01/27/2025 | N | Υ |
| Holbrook Kathryn Data Collection SP N N RN P N 12/12/2018 Y 03/09/2021 N N | Hawthorne | James | Medical Supervisor | SP | N | N | MD | Р | Υ | 05/09/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| | Hays | Lon | Medical Supervisor | SP | N | N | MD | Р | Υ | 11/08/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| Humphrice Tiresthy Date Collection CD N N DN D V 00/04/0000 V V | Holbrook | Kathryn | Data Collection | SP | N | N | RN | Р | N | 12/12/2018 | | Υ | 03/09/2021 | N | N |
| Tumprines filliothy Data Collection SP N N KN P Y 02/21/2023 Y Y 01/23/2025 N Y | Humphries | Timothy | Data Collection | SP | Ν | N | RN | Р | Υ | 02/21/2023 | Υ | Υ | 01/23/2025 | N | Υ |

| | | | | | | | | | | | | | 331 | 70 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Last Name | First Name | Responsibility In<br>Project | Role | A<br>C | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | Last<br>Updated | SFI | Active |
| Hurt | Amber | Data Collection | SP | Υ | N | | Р | N | 06/14/2021 | | Υ | 06/15/2022 | N | Υ |
| Islam | Mohammed | Medical Supervisor | SP | N | N | MD | Р | Υ | 10/12/2023 | Υ | Υ | 01/27/2025 | Ν | Υ |
| Jackson | Kayleigh | Data Collection | SP | N | N | CNA | Р | N | 10/31/2017 | | Υ | 10/14/2020 | N | N |
| Jones | Dowana | Data Collection | SP | N | N | | Р | N | 04/18/2021 | | Υ | 04/29/2022 | Ν | Υ |
| Knight | Stephanie | Data Collection | SP | N | N | RN | Р | N | 10/20/2020 | | Υ | 04/29/2022 | N | Υ |
| Kroupa | Spencer | Data Collection | SP | N | N | | | Υ | 06/07/2023 | Υ | Υ | 06/17/2024 | N | N |
| Kunzelman | Wyatt | Data Collection | SP | Υ | N | | | Υ | 09/12/2023 | Υ | Υ | 01/21/2025 | N | N |
| Lester | Clark | Medical Supervisor | SP | N | N | MD | Р | N | 07/05/2022 | Υ | Υ | 01/27/2025 | N | Υ |
| Leung | Steve | Medical Supervisor | SP | N | N | MD | Р | Υ | 10/01/2024 | Υ | Υ | 01/27/2025 | N | Υ |
| Lewis | Russell | Data Collection | SP | Υ | N | ВА | Р | N | 02/16/2021 | | Υ | 09/08/2022 | N | N |
| Long | Konnor | Data Collection | SP | Υ | N | | Р | N | 06/20/2019 | | Υ | 06/24/2020 | N | N |
| Mandal | Anjana | Data Collection | SP | N | N | | S | N | 12/22/2021 | Υ | Υ | 01/21/2025 | N | Υ |
| Mandal | Prabin | Data Collection | SP | N | N | | | N | 06/27/2022 | Υ | Υ | 06/17/2024 | N | N |
| Mann | Shannon | Data Collection | SP | N | N | RN | Р | N | 01/21/2021 | | Υ | 11/30/2021 | N | N |
| Maynard | Marshall | Data Collection | SP | N | N | | Р | N | 06/16/2022 | Υ | Υ | 06/17/2024 | N | N |
| McClanahan | Sarah | Medical Supervisor | SP | N | N | MD | Р | Υ | 02/17/2023 | Υ | Υ | 01/27/2025 | N | Υ |
| McGee | Paul | Data Collection | SP | Υ | N | | Р | Υ | 04/25/2025 | Υ | Υ | 08/20/2025 | N | Υ |
| Meadows | Amy | Medical Supervisor | SP | N | N | MD,<br>MHS,<br>FAA | Р | Υ | 09/27/2024 | Υ | Υ | 01/27/2025 | N | Υ |
| Milward | Brenda | Project Assistance/Support | DP | Υ | N | | Р | N | 04/10/2019 | | Υ | 06/24/2020 | N | N |
| Min | James | Medical Supervisor | SP | N | N | MD | Р | Υ | 10/23/2023 | Υ | Υ | 01/27/2025 | N | N |
| Minix | Kathleen | Data Collection | SP | N | N | RN | Р | N | 04/12/2021 | | Υ | 04/29/2022 | N | Υ |
| Nadim | Amina | Project Assistance/Support | SP | N | N | | S | N | 02/16/2021 | Υ | Υ | 06/14/2022 | N | Υ |
| Nanda | Jassimran | Data Collection | SP | N | N | | P | N | 01/07/2019 | | Υ | 06/24/2020 | N | N |
| Napier | Janice | Data Collection | SP | N | N | RN | P | N | 10/27/2020 | Υ | Y | 06/28/2023 | N | N |
| Neltner | Matthew | Medical Supervisor | SP | N | N | MD | P | Υ | 03/11/2024 | Y | Υ | 03/05/2021 | N | Υ |
| Nichols | Jocelyn | Data Collection | SP | Υ | N | | P | N | 07/24/2019 | | Y | 06/24/2020 | N | N |
| Nieto | Alayne | Data Collection | SP | N | N | RN | P | Y | 04/18/2025 | Υ | Y | 01/23/2025 | N | Y |
| Oller | Devin | Consultant/Advisor | SP | N | N | | | Y | | Y | Υ | 08/20/2025 | N | N |
| Oros | Sarah | Medical Supervisor | SP | N | | MD | P | Y | 02/16/2023 | Y | Y | 01/27/2025 | N | Y |
| Parson | Lee | Data Collection | SP | N | N | RN | P | Y | 07/03/2024 | Y | Y | 01/23/2025 | N | Y |
| Potter | Samuel | Medical Supervisor | SP | N | | MD | P | Y | 01/06/2023 | Y | Y | 01/27/2025 | N | Y |
| Quarles | Allison | Data Collection | SP | N | N | RN | P | Y | 11/12/2024 | Y | Y | 01/23/2025 | N | Y |
| Rakesh | Gopalkumar | Medical Supervisor | SP | N | N | MD | P | Y | 09/15/2022 | Y | Y | 01/27/2025 | N | Υ |
| Rayapati | Abner | Medical Supervisor | SP | N | N | MD | P | N | 04/19/2021 | Y | Y | 06/28/2023 | N | N |
| Rice | Linda | Data Collection | SP | N | N | RN, | Р | Y | 11/14/2024 | Y | Y | 04/29/2022 | N | N |
| | | | | | | CCRC | | | | | | | | Υ |
| Roads | Andrew | Medical Supervisor | SP | N | N | MD | Р | N | 05/11/2022 | Y | Y | 10/04/2021 | N | |
| Rogers | Karen | Data Collection | SP | N | N | RN | Р | Y | 01/15/2025 | Y | Y | 01/23/2025 | N | Y |
| Ross | Dorothy | Data Collection | SP | N | N | CRA | Р | Y | 11/03/2023 | Y | Y | 01/23/2025 | N | Y |
| Rudd | Triana | Data Collection | SP | N | N | | Р | N | 09/16/2021 | Y | Y | 02/01/2024 | N | N |
| Rudd | Trinity | Data Collection | SP | N | N | DN | Р | N | 09/22/2020 | Y | Y | 06/28/2023 | N | N |
| Rusch | Kali | Data Collection | SP | N | N | RN | Р | Y | 07/12/2024 | Y | Y | 01/23/2025 | N | Y |
| Shelton | Charles | Medical Supervisor | SP | N | N | MD | Р | Y | 04/05/2023 | Υ | Y | 01/27/2025 | N | Y |
| Shraberg | David | Medical Supervisor | SP | N | N | MD | Р | N | 10/16/2018 | | Y | 10/14/2020 | N | N |
| Silverstein | Lily | Data Collection | SP | N | | RN | S | Y | 11/30/2024 | Y | Y | 02/01/2024 | N | Y |
| Skaggs | Kylee | Data Collection | SP | N | N | RN | Р | Y | | Y | Y | 10/18/2022 | N | Y |
| Sloan | Paul | Medical Supervisor | SP | N | | MD | Р | Y | | Υ | Y | 01/27/2025 | N | Y |
| Smith | Kayla | Data Collection | SP | N | N | | Р | N | 06/04/2019 | | Υ | 10/05/2021 | N | N |

| Last Name | First Name | Responsibility In<br>Project | Role | A<br>C | Contact | Degree | StatusFlag | (HSP) | (HSP)Date | (RCR) | Removed? | Last<br>Updated | SFI | Active |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Smoot | Holly | Data Collection | SP | N | N | RN | Р | N | 08/17/2021 | | Υ | 04/29/2022 | N | N |
| Stamper | Brady | Data Collection | SP | N | N | | Р | Υ | 06/05/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Stanley | Catherine | Data Collection | SP | Υ | N | | Р | N | 05/11/2021 | Υ | Υ | 02/03/2023 | N | Ν |
| Stephens | Tonya | Data Collection | SP | N | N | RN | Р | Υ | 08/16/2025 | Υ | Υ | 09/04/2024 | N | Υ |
| Stiehler | Julie | Data Collection | SP | N | N | RN | Р | Υ | 05/29/2024 | Υ | Υ | 04/29/2022 | N | Υ |
| Swain | Audrie | Data Collection | SP | N | N | | Р | Υ | 02/11/2025 | Υ | Υ | 01/23/2025 | N | Υ |
| Tarr | Rebecca | Project<br>Assistance/Support | SP | N | N | RN | Р | N | 10/08/2020 | Υ | Υ | 06/28/2023 | N | Υ |
| Tarrence | Jacob | Data Collection | SP | Υ | N | | Р | N | 04/20/2021 | | Υ | 10/04/2021 | N | N |
| Taylor | Cinnamon | Data<br>Analysis/Processing | SP | N | N | | S | N | 01/14/2019 | | Υ | 06/24/2020 | N | N |
| Telfair Hull | Alexandra | Data Collection | SP | N | N | | Р | N | 02/26/2019 | | Υ | 10/14/2020 | N | N |
| Thompson | Tamra | Data Collection | SP | Υ | N | | | Υ | 09/28/2022 | Υ | Υ | 09/06/2024 | N | N |
| Tillery | Melanie | Data Collection | SP | N | N | RN | Р | Υ | 09/05/2024 | Υ | Υ | 06/14/2022 | N | Υ |
| True | Laura | Data Collection | SP | N | N | | Р | N | 04/13/2020 | | Υ | 06/14/2022 | N | N |
| Tuttle | Teresa | Data Collection | SP | N | N | RN | Р | Υ | 02/25/2023 | Υ | Υ | 01/23/2025 | N | Υ |
| Vincent | Sylvia | Data Collection | SP | N | N | | Р | Υ | 01/30/2024 | Υ | Υ | 01/21/2025 | N | Υ |
| Watts | Linda | Data Collection | SP | N | N | RN | Р | N | 11/10/2021 | Υ | Υ | 02/01/2024 | N | N |
| Wengert | Brandon | Recruitment | SP | N | N | | Р | Υ | 01/15/2025 | Υ | Υ | 07/07/2021 | N | Υ |
| White | Jessica | Data Collection | SP | N | N | RN | Р | Υ | 02/23/2023 | Υ | Υ | 09/04/2024 | N | N |
| Wilmhoff | Jenna | Data Collection | SP | N | N | RN | Р | Υ | 07/02/2024 | Υ | Υ | 01/23/2025 | N | Υ |
| Wilson | Aimee | Data Collection | SP | N | N | RN | Р | N | 06/22/2022 | Υ | Υ | 10/18/2022 | N | N |
| Woodson | Andrea | Data Collection | SP | Υ | N | RN | Р | N | 05/13/2021 | | Υ | 09/07/2022 | N | N |
| Yadon | Rachele | Medical Supervisor | SP | N | N | MD | Р | Υ | 01/09/2025 | Υ | Υ | 01/27/2025 | N | Υ |
| Young | Cherish | Data Collection | SP | N | N | CNA | Р | Υ | 11/23/2024 | Υ | Υ | 03/13/2020 | N | Υ |
| Zeidan | Ronnie | Medical Supervisor | SP | Ν | N | MD | S | N | 07/11/2018 | | Υ | 10/14/2020 | N | N |

#### RESEARCH DESCRIPTION

0 unresolved comment(s)

You may attach a sponsor's protocol pages in the "Additional Information" section and refer to them where necessary in the Research Description. However, each prompt that applies to your study should contain at least a summary paragraph.

#### Pro Tips:

- . Save your work often to avoid losing data.
- Use one of the attachment buttons in this section or under the Additional Information section to include supplemental
  information with your application. During the document upload process, you will be able to provide a brief description
  of the attachment.

#### **Background**

Include a brief review of existing literature in the area of your research. You should identify gaps in knowledge that should be addressed and explain how your research will address those gaps or contribute to existing knowledge in this area. For interventional research, search PubMed and ClinicalTrials.gov for duplicative ongoing and completed trials with same condition and intervention(s).

Despite the known risks of co-administration of opioids and alcohol and admonitions against their co-administration in product package inserts, the two are commonly used in combination. Very few controlled studies have examined the nature of the interaction between oxycodone/opioids and ethanol. One study examined drug naïve individuals and tested two doses of ethanol (0.3 and 0.6 g/kg) in combination with a single therapeutic dose of oxycodone (10 mg) (Zacny et al., 2011). That report indicated that neither the low dose of ethanol nor of oxycodone produced subjective reports related to abuse liability alone but did so when combined. A second study examined hydromorphone (1 and 2 mg) in combination with alcohol and concluded that hydromorphone did not alter alcohol's pharmacodynamic effects (Rush, 2001). Both of these studies tested relatively low doses of opioids and enrolled non-experienced opioid users. A third study reported no additive or interaction effects and no pharmacokinetic interactions of morphine (50 mg) with a single dose of ethanol (0.7 g/kg) (Setnik et al., 2014). Subsequent re-randomization of the moderate-drinking male-only cohort to either a lower (30 mg) or higher (80 mg) morphine dose still produced no interactions. Another study, and perhaps the most relevant, reported that IV ethanol enhanced oxycodone (20 mg) -induced hypercapnia (van der Schrier et al., 2017). These studies are collectively informative; however, none of these studies fully examined a dose response relationship or enrolled individuals who combine opioids and alcohol as part of their drug use pattern as will be done in the proposed study.

#### **Objectives**

List your research objectives. Please include a summary of intended research objectives in the box below.

- 1. Characterize the physiological response and subjective profile of oxycodone
- 2. Characterize the physiological response and subjective profile of alcohol
- 3. Assess the acute physiological response and subjective profile to oxycodone and alcohol combinations

## **Study Design**

Describe and explain the study design (e.g., observational, secondary analysis, single/double blind, parallel, crossover, deception, etc.).

- Clinical Research: Indicate whether subjects will be randomized and whether subjects will receive any placebo.
- Community-Based Participatory Research: If you are conducting community-based participatory research (CBPR), describe
  strategies for involvement of community members in the design and implementation of the study, and dissemination of results from
  the study.
- Qualitative research: Indicate ranges where flexibility is needed, if a fixed interview transcript is not available, describe interview
  topics including the most sensitive potential questions.
- Research Repositories: If the purpose of this submission is to establish a Research Repository (bank, registry) and the material
  you plan to collect is already available from a commercial supplier, clinical lab, or established IRB approved research repository,
  provide scientific justification for establishing an additional repository collecting duplicate material. Describe the repository design
  and operating procedures. For relevant information to include, see the <a href="UK Research Biospecimen Bank Guidance">UK Research Registry Guidance</a>.

An initial pilot study will employ a quasi-randomized, double-blind, placebo-controlled, inpatient, within-subjects design. Doses of oxycodone alone and alcohol alone will be given in random order. In regard to the dose combinations, during the pilot study subjects will receive 20 mg Oxy + 0.5 g/kg ETOH as the first combination dose and 40 mg OXY + 0.8 g/kg ETOH as the last combination dose. The purpose of this constrained (i.e., quasi-randomized) approach is to ensure that all dose combinations are safely tolerated. Between 3-6 volunteers will complete the pilot phase, and a review of safety will be conducted. Findings will be shared with the IRB for approval to proceed to the fully randomized phase of the study.

After completion of the pilot phase study, a fully randomized, double-blind, placebo-controlled, inpatient, within-subjects design will be utilized.

| Attach Type | File Name |
|-------------|---------------------------------------------------------|
| StudyDesign | Opioids & Alcohol Pilot Phase Completion 2-14-2023.docx |

#### **Subject Recruitment Methods & Advertising**

Describe how the study team will identify and recruit subjects. Please consider the following items and provide additional information as needed so that the IRB can follow each step of the recruitment process.

- How will the study team identify potential participants?
- Who will first contact the potential subjects, and how?
- Will you use advertisements? If so, how will you distribute those?
- How and where will the research team meet with potential participants?
- If applicable, describe proposed outreach programs for recruiting women, minorities, or disparate populations.
- How you will minimize undue influence in recruitment?
- Attach copies of all recruiting and advertising materials (emails, verbal scripts, flyers, posts, messages, etc.).

For additional information on recruiting and advertising:

- IRB Application Instructions Advertisements
- Pl Guide to Identification and Recruitment of Human Subjects for Research

Volunteers will be recruited via the advertising methods listed below (Advertising) and will make initial contact by phone, BuildClinical, or Facebook with one of our staff who have completed the research training and HIPAA compliance web-based teaching modules. If the volunteer discloses information that would make him/her potentially eligible for the study, they will be invited to come in for a screening appointment. Screening is completed by one of our trained research assistants/research nurses/investigators at the Straus Behavioral Science Research Building or the UK CCTS. Study investigators may interact with volunteers in any of these settings and appropriate precautions are in place to ensure privacy during the intake process.

Volunteers will be recruited through newspaper and radio advertisement, local postings, online advertisements on forums such as ResearchMatch, BuildClinical, Facebook, Craigslist, by geo-fencing techniques (advertising within a defined geographical location) and by word-of-mouth. Our Facebook page template and study flyers have been approved by UK PR.

## Attachments

| Attach Type | File Name |
|-------------|----------------------------------------------------------|
| Advertising | Opioid & Alcohol ads (clean).pdf |
| Advertising | Possible Accompanying Text for Online Ads APPROVED.pdf |
| Advertising | 20201 Op x alcohol PR approved ads - 03.20.2020.pdf |
| Advertising | Facebook page - revised Dec 17 APPROVED.pdf |
| Advertising | BuildClinical Landing Page - PR stamped.pdf |
| Advertising | BuildClinical Opioid ads - PR stamped.pdf |
| Advertising | BuildClinical Secure questionnaire.pdf |
| Advertising | Tracked Changes - BuildClinical Secure questionnaire.pdf |
| Advertising | Opioid & Alcohol Flyer 6.8.22 (CLEAN).pdf |
| Advertising | Opioid & Alcohol - Cards 6.8.22 (CLEAN).pdf |
| Advertising | Opioid & Alcohol - Cards 6.8.22 (PR Approved).pdf |
| Advertising | Opioid & Alcohol Flyers 6.8.22 (PR APPROVED).pdf |
| Advertising | Opioid & Alcohol - Digital ads 6.8.22 (PR APPROVED).pdf |
| Advertising | Opioids & Alcohol Digital Ads 6.8.22 (CLEAN).pdf |

#### **Research Procedures**

Describe how the research will be conducted.

- What experience will study participants have?
- · What will study participants be expected to do?
- How long will the study last?
- Outline the schedule and timing of study procedures.
- Provide visit-by-visit listing of all procedures that will take place.
- Identify all procedures that will be carried out with each group of participants.
- Describe deception and debrief procedures if deception is involved.

Differentiate between procedures that involve standard/routine clinical care and those that will be performed specifically for this research project. List medications that are explicitly forbidden or permitted during study participation.

Screening and Admission: Subjects will answer questionnaires related to their drug use and health during screening. They will also undergo medical examination that includes a physical exam, electrocardiogram (ECG), and blood and urine chemistries. The number of screening visits may vary depending on the subjects' availability and staff scheduling. This study will enroll only non-physically-dependent, recreational alcohol/opioid users who have prior non-medical experience with both opioids and alcohol in the past year; supervised urine samples must corroborate self-reports. Female participants will be tested at screening, on entry, at weekly intervals, and prior to each session for pregnancy. Prior medical records may be obtained with volunteer consent if there is any question about the volunteers' health history. Each participant will sign a form that details the HIPAA-compliant manner in which research material is collected.

During screening, each subject will complete a cold pressor test (CPT), which will be performed during the main study (see description below). Subjects that are unable to tolerate the CPT or who report no pain during the CPT will be excluded from the study.

General Methods: After admission to the inpatient unit, a trained research staff person will familiarize the participant with the various computer tasks to ensure that they are comfortable with the tasks prior to study initiation. All experimental session procedures will be conducted with methods that have been previously used to study the effects of psychoactive drugs. Some physiological measures (e.g., heart rate, resting blood pressure, and oxygen saturation) will be collected using a Macintosh computer system that is interfaced with physiological monitoring equipment (DINAMAP) and will be monitored continuously throughout the sessions. Other physiological measures (e.g., respiratory rate) will be collected at regular intervals. These measures serve as both safety data and as study outcomes. An array of subjective and observer-rated measures, including but not limited to visual analog scales and Likert adjective checklists, are presented on a computer screen and a computer mouse is used to respond to questions. CPT will be used to measure analgesia. Smoking is allowed at any time with an escort, though only under supervised conditions, with the exception of 30 minutes prior to the start of the session and until the session is completed. A trained research staff will be present throughout the entire session.

Experimental Procedures: Prior to starting the experiment, subjects will participate in an initial active control test session during which the subjects will receive 30 mg oxycodone (oral). This session will serve as a "qualifying day" or responsiveness challenge which is intended to confirm that subjects are able to detect the active drug and report "liking" for the test agent (i.e., confirmation that the subject will provide a sensitive signal). If subjects fail to report any drug liking and identify the drug as placebo, they may not proceed further with dosing.

Experimental Sessions: During each session, subjects will receive two oral doses. All dosing will be double dummy – subjects will always receive one capsule preparation (oxycodone or placebo) and one liquid preparation (alcohol [ETOH] or placebo). A total of ten [including the active control test session described above] 6.5 hr sessions will be conducted including 30 min of baseline data collection. Dose conditions will include: 0 mg OXY & 0 g/kg ETOH, 20 mg OXY & 0 g/kg ETOH, 40 mg OXY & 0 g/kg ETOH, 0 mg OXY & 0.5 g/kg ETOH, 40 mg OXY & 0.8 g/kg ETOH, 20 mg OXY & 0.5 g/kg ETOH, 20 mg OXY & 0.8 g/kg ETOH. Due to differences in body fat, alcohol doses will be decreased by 15% for women. Sessions will be at least 48 hrs apart to ensure adequate wash-out. Dosing will be staggered in order to align their peak responses (Tmax). The reported Tmax for oxycodone is estimated at ~1.5 hr and for alcohol is ~1 hr; therefore, oxycodone will be administered 0.5 hr before alcohol.

Discharge & Follow-up Appointment: Subjects will typically be discharged from the CCTS the day after they complete their final session. They may be discharged early for safety reasons (see below) or if they fail to comply with the protocol or the inpatient rules (e.g. verbal abuse of staff). They will be asked before they leave if they are interested in treatment for their substance abuse and offered referrals for treatment if they indicate interest. A follow-up appointment will be scheduled within two weeks of discharge. The volunteers will be asked about their health status, drug use, and any adverse events occurring since discharge. The follow-up appointment may be conducted over the phone or in person at the Robert Straus Behavioral Research Facility.

## Attachments

#### **Data Collection & Research Materials**

In this section, please provide the following:

• Describe all sources or methods for obtaining research materials about or from living individuals (such as specimens, records, surveys, interviews, participant observation, etc.), and explain why this information is needed to conduct the study.

- For each source or method described, please list or attach all data to be collected (such as genetic information, interview scripts, survey tools, data collection forms for existing data, etc.).
- If you will conduct a record or chart review, list the beginning and end dates of the records you will view.

During the screening phase of the study, data collected will include demographics, medical history, NEO, drug use history, results of laboratory tests (blood and urine chemistries and ECG), and results of urine drug screens.

Outcome measures collected during the inpatient phase of the study include physiological measures (e.g., pupil diameter, expired CO2, blood pressure, heart rate, respiration rate, breath alcohol concentration), subject-rated questionnaires (e.g., Visual Analog Scales for drug effects, Pharmacological Class Questionnaire, Street Value Questionnaire, Next-Day Questionnaire), responses to the Cold Pressor Test, observer ratings, and psychomotor/cognitive tasks (such as the Digit Symbol Substitution Task, and the Balance Task, Circular Lights task, and Flicker Fusion Task: descriptions of these tasks are below).

The Circular Lights Task: The circular lights task involves rapid hand-eye coordinated movements in which a participant presses a series of 16 buttons (circularly arranged around a 54-cm diameter) as rapidly as possible in response to the randomly sequenced illumination of their associated lights. Score equals the number of correct button presses in a 60-sec trial.

The Digit Symbol Substitution Task: The representation of a 9-key keypad is illustrated on a computer screen. Each trial illustrates a randomly selected pattern with one position illuminated in each of the three horizontal key rows. Subjects press button positions on the computer keypad to reproduce the pattern on screen. The number of trials attempted, the number of correct trials, and the percentage of correct trials during the 90-sec test period are scored.

The Balance Task: This task assesses the participant's ability to stand upright on one foot with eyes closed and arms extended to the side at shoulder height (for a maximum of 30 seconds on each foot).

The Flicker Fusion Task: The Flicker Fusion task is used widely to detect the sedative properties of various drug classes, including opioids, antihistamines, benzodiazepines and barbiturates. It provides a sensitive assessment of integrated CNS processing and attention and is sensitive to changes in cortical arousal. A red-light stimulus flickers at varying frequencies. The frequency at which the subject identifies the light as no longer flickering (i.e., a continuous light signal) is the critical fusion frequency (as the frequency increases) and the frequency at which the subject identifies the light as flickering after fusion (as the frequency decreases) is the critical flicker frequency.

## Attachments

| Attach Type File Name | |
|---|---|
| DataCollection | Screening Questionnaires - 03.20.2020.pdf |
| DataCollection | Session Questionnaires - 03,20,2020.pdf |

#### Resources

Describe the availability of the resources and adequacy of the facilities that you will use to perform the research. Such resources may include:

- Staffing and personnel, in terms of availability, number, expertise, and experience;
- Computer or other technological resources, mobile or otherwise, required or created during the conduct of the research;
- Psychological, social, or medical services, including equipment needed to protect subjects, medical monitoring, ancillary care, or counseling or social support services that may be required because of research participation;
- Resources for communication with subjects, such as language translation/interpretation services.

The study will take place at our laboratory and at the University of Kentucky CCTS Inpatient Unit. Screening procedures will largely be performed at our laboratory while enrolled patients will perform experimental procedures and reside at the CCTS. Experimental rooms at the CCTS are equipped with the necessary physiologic and computer equipment necessary for the study. There will be 24- hr nursing supervision of volunteers while in the hospital. Dr. Michelle Lofwall will be the primary medically responsible investigator and is an adult psychiatrist with ACLS certification who has worked extensively with individuals with substance use disorders both in clinical and research settings. The Psychiatry Attending Service will monitor subjects daily while they are inpatients. Dr. Walsh will provide oversight for the study. Overall, the study team and the resources described above are well equipped to protect the participants and successfully implement, carry out, and complete this study protocol.

#### **Potential Risks & Benefits**

#### Risks

- Describe any potential risks including physical, psychological, social, legal, ability to re-identify subjects, or other risks. Assess the seriousness and likelihood of each risk.
- Which risks may affect a subject's willingness to participate in the study?
- Describe likely adverse effects of drugs, biologics, devices or procedures participants may encounter while in the study.
- Qualitative research describe ethical issues that could arise while conducting research in the field and strategies you may use to handle those situations.
- Describe any steps to mitigate these risks.

#### **Benefits**

- Describe potential direct benefits to study participants including diagnostic or therapeutic, physical, psychological or emotional, learning benefits. This cannot include incentives or payments.
- State if there are no direct benefits.

Describe potential benefits to society and/or general knowledge to be gained.

Describe why potential benefits are reasonable in relation to potential risks. If applicable, justify why risks to vulnerable subjects are reasonable to potential benefits.

The primary risks for the subjects in this study are associated with drug administration. Typical side effects of oxycodone include nausea, vomiting, headache, dry mouth, itchiness, drowsiness, sweating, dizziness, stimulation, somnolence, lightheadedness, restlessness, euphoria, talkativeness, urinary retention, and constipation. More serious side effects may include allergic reaction and respiratory depression, but these are rare and unlikely to occur in a sample of volunteers who have experience using opioids illicitly. Side effects of alcohol include: somnolence, vomiting, diarrhea, nausea, headache, blurred vision, slurred speech, and difficulty breathing. We have carefully chosen doses to minimize serious drug effects. The combination of these two drugs may have additive or synergistic effects, but doses have been carefully selected and safety will be carefully monitored (see below).

During the screening process, it is possible that subjects may feel uncomfortable answering personal questions about their health, psychiatric, and drug use histories. However, they may stop answering questions at any point (and are informed of this option during the informed consent process). Participants will have blood drawn via venipuncture, which may cause soreness, bruising, pain, infection, possible fainting, and/or bleeding. Using sterile procedures and well-trained staff minimizes these risks. There is the risk that someone other than the research staff may see a subject's Protected Health Information.

The cold water task produces some painful sensations. However, the participant has full control over their exposure and can remove their arm from the cold water at any point during the trial. The safety cut-off of 5 minutes of immersion was selected to avoid the risk of tissue damage. We have successfully and safely used this model in several other studies without any safety concerns. There are no direct benefits to volunteers. There are potential indirect benefits to society including the knowledge regarding safety, abuse liability, and pharmacodynamics of oxycodone and alcohol (two often co-abused drugs) alone and in combination. Volunteers will indirectly benefit from receiving a free medical evaluation and free meals. If subjects decide they would like substance abuse treatment during the course of the study, we will assist them in finding treatment programs and getting them on the appropriate waiting lists. The amount of risk to which individual study volunteers are exposed to is low. Overall, the risk/benefit ratio appears favorable, and the conduct of this research seems well justified.

#### **Available Alternative Opportunities/Treatments**

Describe alternative treatments or opportunities that might be available to those who choose not to participate in the study, and which offer the subject equal or greater advantages. If applicable, this should include a discussion of the current standard of care treatment(s).

This is not a treatment study. If volunteers express interest in treatment, they will be given referrals and not allowed to participate in this study.

Back to Top

## Records, Privacy, and Confidentiality

Specify where the data and/or specimens will be stored and how the researcher will ensure the privacy and confidentiality of both. Specify who will have access to the data/specimens and why they need access.

Describe how data will be managed after the study is complete:

- If data/specimens will be maintained, specify whether identifiers will be removed from the maintained information/material.
- If identifiers will not be removed, provide justification for retaining them and describe how you will protect confidentiality.
- If the data/specimens will be destroyed, verify that this will not violate <u>retention policies</u> and will adhere to applicable facility requirements.

If this study will use de-identified data from another source, describe what measures will be taken to ensure that subject identifiers are not given to the investigator.

If applicable, describe procedures for sharing data/specimens with collaborators not affiliated with UK.

For additional considerations:

Return of Research Results or Incidental Research Findings

**HIPAA** policies

**FERPA policies** 

Procedures for Transfer agreements

Information regarding multi-site studies

NIH Genomic Data Sharing (GDS) Policy

Digital Data

Sources of research material obtained from our volunteers during screening and study participation include: blood and urine specimens, expired breath samples for alcohol, ECG data, self-reported information on physical and mental health, family history, drug and alcohol use history, demographic information, volunteer and study staff observation of drug effects, vital signs (e.g. temperature, blood pressure, heart rate), and other physiological measures. All this information is required to determine eligibility for the study, to ensure safety during the experimental sessions and for outcome measures. All research material will be obtained and discarded when necessary in a HIPAA-complaint manner. All materials will be collected specifically for the proposed study by trained staff. The

principal investigator and medical team will have access to private health information about volunteers so that study eligibility can be determined. All data with personal health information are kept in a locked file cabinet that is separate from a locked file cabinet with deidentified volunteer data. Prior medical records may be obtained with volunteer consent if there is any question about the volunteers' health history. Each participant will sign a form that details the HIPAA-compliant manner in which research material is collected.

If in the course of the research study, the investigators discover something that could affect the health of a subject, the medical monitor will determine if it is in the best interest of the subject to disclose the finding. If the information is to be disclosed, a trained member of the research team or the medical monitor will inform the subject of the finding and advise them to follow up with a primary care doctor or other appropriate entity.

Identifying information will be stored in a separate locked file cabinet from all other data and codes that could link an individuals' Subject ID to their identity. Incidental materials containing subject identifiers will be shredded or incinerated. Electronic data will be stored on password-protected computers in password-protected files. Access to identifying information will only be available to key research personnel. In addition, a Certificate of Confidentiality will be obtained. Biological samples will be destroyed no later than after study completion but typically soon after discharge. Paper records will be locked and stored for a minimum of 7 years and destroyed through shredding or a professional destruction company.

Subjects will be carefully screened (history and physical examination, routine labs including CBC and LFTs, urinalvsis. ECG. and psychiatric assessments) to exclude those with a risk of adverse events. Those at increased risk may have histories that include a personal or family history of seizure or head injury associated with more than a brief loss of consciousness, hypertension, psychosis, etc. During sessions, subjects remain under careful observation. Vital signs will be collected multiple times daily throughout the dosing period. Dr. Walsh has substantial experience in testing psychoactive substances in human subjects. Female subjects will be given pregnancy tests weekly and before each session to ensure that we do not administer any potentially harmful agents to a pregnant woman. To protect confidentiality, all research subjects are identified by a subject identification code (Subject ID) consisting of their initials and sequentially assigned subject numbers on all forms and data files, and not by their names. Actual subject names and corresponding subject IDs are kept in a locked master file separate from the actual data collected during the study. All personal and experimental information is kept locked and is accessible only to key personnel involved in the research. Risks of allergic reaction or serious respiratory depression are mitigated by the volunteer histories of opioid use. However, should an allergic reaction occur, diphenhydramine will be available for oral administration. During test sessions when opioids are administered, if respiratory rate drops below 10 breaths/min accompanied by sedation, volunteers are verbally prompted to breathe. In our experience, physical (e.g., gentle shaking) and verbal stimulation is often sufficient to prompt breathing and restore a normal respiratory rate. During test sessions, nurses are instructed to check and record oxygen saturation and respiratory rate before each drug administration as follows: If respiratory rate falls below 10 breaths/min or oxygen saturation is less than 95%, REPEAT and count breaths for 60 seconds. If either oxygen saturation or respiratory rate remains outside parameters, HOLD the study medication and call the study physicians. If the patient is unresponsive, call code team. Naloxone and supplemental oxygen may be administered based on physician evaluation. If oxygen saturation falls below 90, any subsequent dosing is terminated and participants remain under continuous monitoring until resolved. The study takes place within a fully functional hospital with emergency code response available. We do not anticipate needing to employ these interventions but they are available in the event of an emergency.

Because we are exploring possible synergistic or additive effects of oxycodone and alcohol, this study includes a quasi- randomized, double-blind, placebo-controlled pilot phase to ensure that all dose conditions are safely tolerated before moving to a fully randomized dose order. Up to six volunteers will participate in the pilot phase, and a full safety assessment will be made in order to determine if dose adjustment is necessary for the full study.

Participants choosing to leave the study early will be advised to complete a vitals check before leaving the research facility (Inpatient Unit, Straus Building). However, we are not permitted to retain participants against their will, so they may choose to leave AMA before a vitals check or before research staff are able to notify to the investigator/physician.

THE policies state that IRB-related research records must be retained for a minimum of 6 years after study closure. Check this item to confirm that you will retain all IRB-related records for a minimum of 6 years after study closure.

#### **Payment**

Describe the incentives (monetary or other) being offered to subjects for their participation. If monetary compensation is offered, indicate the amount and describe the terms and schedule of payment. Please review this guidance for more information on payments to subjects, including restrictions and expectations.

Participants will be paid for each screening visit at the rate of \$50/visit. If only a urinalysis is required, subjects will be paid \$15.

For the main inpatient study phase, participants will receive a base pay of \$60/night regardless of whether or not they complete the study. They will receive a bonus of \$60/night if they complete the entire study, but not in the case of early departure or dismissal. If the volunteer completes the study, depending on their length of stay, they may receive a maximum of approximately \$3,600 (for 30 study nights). This is consistent with the current compensation for similar studies.

There will be one follow up appointment after discharge from the inpatient unit, and individuals will be paid \$25 for this visit.

Travel reimbursement will be available to participants (up to \$60) based on location. Participants traveling from Fayette county will not be reimbursed for travel. Participants traveling from Scott, Bourbon, Clark, Woodford, Jessamine, or Madison county will be reimbursed \$12 for travel. Participants traveling from Grant, Harrison, Nicholas, Bath, Montgomery, Powell, Estill, Garrard, Mercer, Anderson, Franklin, or Owen county will be reimbursed \$23 for travel. Participants traveling from Boone, Kenton, Campbell, Pendleton, Bracken, Robertson, Mason, Fleming, Rowan, Menifee, Wolfe, Lee, Owsley, Jackson, Rockcastle, Laurel, Pulaski, Lincoln, Casey,

Boyle, Washington, Marion, Nelson, Spencer, Shelby, Henry, Carroll, or Gallatin county will be reimbursed \$45. Participants traveling from Kentucky counties not listed above or from out of state will be reimbursed \$60 for travel.

Participants will be paid in \$500 increments. They will be given their first payment at discharge. We will mail them the remainder of the checks. We will mail them \$500 per check per day until they are fully paid. We will mail the checks to the address that they provide us. Alternatively, participants are permitted to visit our office to pick up checks in-person during normal business hours Monday-Friday. This method of payment has been previously approved under IRB #47055.

## **Costs to Subjects**

Include a list of services and/or tests that will not be paid for by the sponsor and/or the study (e.g., MRI, HIV). Keep in mind that a subject will not know what is "standard" – and thus not covered by the sponsor/study – unless you tell them.

There will be no cost to volunteers for participation in the current study. Cost of research-related harm will be the subjects' responsibility.

#### **Data and Safety Monitoring**

The IRB requires review and approval of data and safety monitoring plans for greater than minimal risk research or NIH-funded/FDA-regulated clinical investigations.

- If you are conducting greater than minimal risk research, or your clinical investigation is NIH-funded, describe your Data and Safety Monitoring Plan (DSMP). Click here for additional guidance on developing a Data and Safety Monitoring Plan.
- If this is a non-sponsored investigator-initiated protocol considered greater than minimal risk research, and if you are planning on using a Data and Safety Monitoring Board (DSMB) as part of your DSMP, <u>click here for additional guidance</u> for information to include with your IRB application.



Medical Safety Monitoring: Volunteers undergo a rigorous screening process to determine their eligibility and safety of their participation. In addition, our well-trained and vigilant research and medical staff, and the carefully considered medication dosing and safety criteria all serve as precautionary measures to ensure the safety of volunteers. The principal investigator, Sharon L. Walsh, Ph.D., will be the primary person responsible for monitoring the safety of this project, executing the DSMP and complying with all reporting requirements. Our medical staff, including Dr. Lofwall and CCTS nursing staff, will conduct careful medical monitoring. We have an experienced anesthesiologist, Kevin Hatton, M.D. consulting on this project as an additional safety precaution. Volunteers will have daily contact with a physician and CCTS nurses while they reside as inpatients. The safety monitoring of each volunteer is discussed on an ongoing basis among medical and scientific staff, including our study statistician, Paul Nuzzo. This process has been successful in protecting volunteers and the integrity of the scientific outcomes. Any minor adverse events will be reviewed and adjudicated by the study team, documented in the subjects' medical charts through progress notes and medical logs along with any intervention required (e.g. headache requiring Tylenol). Any severe adverse events, whether study related or not, will be reported to the UK IRB and the FDA within 24 hours or as required.

Data Monitoring: Data are collected using a computerized data collection and management system, which eliminates data entry errors. Data files for experimental tasks and physiological measures from each experimental session will be manipulated and combined into a single electronic spreadsheet for each volunteer that can then be used for analysis. Any data manipulation is conducted twice and compared with the original manipulation to ensure accuracy. Research assistants will minimize missing data and adjust potential data collection errors based upon paper questionnaires. All data requiring hand entry (e.g., urinalysis results, pupil diameter) will be double entered by two separate staff members and comparison macros conducted to ensure accuracy. The data are stored on password-protected computers in password-protected files. Data files do not contain PHI. A computer file linking the unique number with the subjects' name will be kept on a stand-alone, password-protected computer available only to the study investigators. All paper copies of the collected data will be stored in locked file cabinets separate from any identifying information. To ensure data integrity and validity, all questionnaires will be explained to volunteers and time for questions and clarifications will be given. Trained research assistants will be present when participants are answering questionnaires to ensure that volunteers are staying on task, paying attention, and to be able to answer any questions from the volunteers should they have questions about the tasks.

**Back to Top** 

#### Future Use and Sharing of Material (e.g., Data/Specimens/Information)

If the material collected for this study will be used by members of the research team or shared with other researchers for future studies, please address the following:

- list the biological specimens and/or information that will be kept
- briefly describe the types, categories and/or purposes of the future research
- describe any risks of the additional use
- · describe privacy/confidentiality protections that will be put into place
- describe the period of time specimens/information may be used
- · describe procedures for sharing specimens/information with secondary researchers
- describe the process for, and limitations to, withdrawal of specimens/data

Investigators may store, use, and share identifiable information for future research. Information will be stored at Robert Straus Behavioral Research Facility for a minimum of 7 years. Investigators will store identifiable information in a password-protected database with access limited to the approved staff. Investigators will remove the participant's name or other direct identifiers and label the information or samples with a code. The key will be stored separately from the master code list. Only select staff will have access to the list that links the code to the individual.

De-identified information may be shared with other researchers without additional consent, provided an IRB has approved this action. If a researcher requests information or samples with identifiable information, an IRB will decide if the research may be conducted with or without consent. Study participants may withdraw permission to allow information or specimen samples to be used for future research via written withdraw request. IRB-approved informed consent outlines this process and provides PI's contact information. Upon receipt of written withdraw request, any remaining specimen samples and information will be destroyed. It may be possible to destroy the code that links the study participant to information or samples. Information and specimen samples that have already been used or shared may not be withdrawn.

Language delineating future use and sharing of research data is already included in IRB-approved consent forms. See Confidentiality section of Research Description for additional information about confidentiality/privacy protections.

Are you recruiting or expect to enroll **Non-English Speaking Subjects or Subjects from a Foreign Culture**? (does not include short form use for incidentally encountered non-English subjects)

○ Yes ○ No

Non-English Speaking Subjects or Subjects from a Foreign Culture

#### **Recruitment and Consent:**

Describe how information about the study will be communicated to potential subjects appropriate for their culture, and if necessary, how new information about the research may be relayed to subjects during the study.

When recruiting Non-English-speaking subjects, provide a consent document in the subject's primary language. After saving this section, attach both the English and translated consent documents in the "Informed Consent" section.

## **Cultural and Language Consultants:**

The PI is required to identify someone who is willing to serve as the cultural consultant to the IRB.

- This person should be familiar with the culture of the subject population and/or be able to verify that translated documents are the equivalent of the English version of documents submitted.
- The consultant should not be involved with the study or have any interest in its IRB approval.
- Please include the name, address, telephone number, and email of the person who agrees to be the cultural consultant for your study.
- ORI staff will facilitate the review process with your consultant. Please do not ask them to review your protocol separately.

For more details, see the IRB Application Instructions on Research Involving Non-English Speaking Subjects or Subjects from a Foreign Culture.

## Local Requirements:

If you will conduct research at an international location, identify and describe:

- · relevant local regulations
- · data privacy regulations
- applicable laws
- · ethics review requirements for human subject protection

Please provide links or sources where possible. If the project has been or will be reviewed by a local ethics review board, attach a copy in the "Additional Information/Materials" section. You may also consult the current edition of the <a href="International Compilation of Human Research Standards">International Compilation of Human Research Standards</a>

Does your study involve HIV/AIDS research and/or screening for other reportable diseases (e.g., Hepatitis C, etc...)? ○ Yes ⓒ No

#### HIV/AIDS Research

If you have questions about what constitutes a reportable disease and/or condition in the state of Kentucky, see ORI's summary sheet: "Reporting Requirements for Diseases and Conditions in Kentucky" [PDF].

**HIV/AIDS Research:** There are additional IRB requirements for designing and implementing the research and for obtaining informed consent. Describe additional safeguards to minimize risk to subjects in the space provided below.

For additional information, visit the online <u>IRB Survival Handbook</u> to download a copy of the "Medical IRB's requirements for Protection of Human Subjects in Research Involving HIV Testing" [D65.0000] [PDF], and visit the <u>Office for Human Research Protections web site</u> for statements on AIDS research, or contact the Office of Research Integrity at 859-257-9428.

## PI-Initiated FDA-Regulated Research

Is this an investigator-initiated study that:

- 1) involves testing a Nonsignificant Risk (NSR) Device, or

## -PI-Sponsored FDA-Regulated Research

If the answer above is yes, then the investigator assumes the regulatory responsibilities of both the investigator and sponsor. The Office of Research Integrity provides a summary list of sponsor IND regulatory requirements for drug trials [PDF], IDE regulatory requirements for SR device trials [PDF], and abbreviated regulatory requirements for NSR device trials [PDF]. For detailed descriptions see FDA Responsibilities for Device Study Sponsors or FDA Responsibilities for IND Drug Study Sponsor-Investigators.

- Describe the experience/knowledge/training (if any) of the investigator serving as a sponsor (e.g., previously held an IND/IDE); and
- Indicate if any sponsor obligations have been transferred to a commercial sponsor, contract research organization (CRO), contract monitor, or other entity (provide details or attach FDA 1571).

This study will be covered under IND # 69,214 (Sponsor: Sharon Walsh, Ph.D.). Dr. Walsh, the Principal Investigator, has been conducting FDA-regulated research for 20+ years. She has held several INDs throughout this period and currently holds three active INDs. She has also served as Principal Investigator for numerous privately sponsored studies in which the IND was held and sponsored by a private company. Through this extensive experience, she is familiar with the submission of INDs, amendments, reporting requirements for adverse events, annual progress reporting requirements and recordkeeping requirements. She is also familiar with Good Clinical Practice guidelines, has participated in numerous related training over the years, and has trained and managed a multi-disciplinary staff on regulatory affairs, confidentiality issues, reporting requirements, data management, data quality assurance, data storage, and human subjects' protections.

IRB policy requires mandatory training for investigators who are also FDA-regulated sponsors (see <u>Sponsor-Investigator FAQs</u>). A sponsor-investigator must complete the applicable Office of Research Integrity web based training, (drug or device) before final IRB approval is granted.

If the sponsor-investigator has completed equivalent sponsor-investigator training, submit documentation of the content for the IRB's consideration.

Attachments
# HIPAA 0 unresolved comment(s)

Is HIPAA applicable? • Yes o No

(Visit ORI's <u>Health Insurance Portability and Accountability Act (HIPAA) web page</u> to determine if your research falls under the HIPAA Privacy Regulation.)



I have attached a HIPAA Waiver of Authorization. c Yes R No

Attachments

#### STUDY DRUG INFORMATION

0 unresolved comment(s)

Drugs are articles intended for use in the diagnosis, cure, mitigation, treatment, or prevention of disease and articles (other than food) intended to affect the structure or any function of the body of man or other animals.

#### The term drug may include:

- · FDA approved drugs,
- unapproved use of approved drugs,
- investigational drugs or biologics,
- other compounds or products intended to affect structure or function of the body, and/or
- <u>complementary and alternative medicine products</u> such as dietary supplements, substances generally recognized as safe (GRAS) when used to diagnose, cure mitigate, treat or prevent disease, or clinical studies of <u>e-cigarettes</u> examining a potential therapeutic purpose.

Does this protocol involve a drug including an FDA approved drug; unapproved use of an FDA approved drug; and/or an investigational drug?

If yes, complete the questions below. Additional study drug guidance.

| Oxycodone, Alcohol | |
|---|---|
| · | |
| Non-Oncology). Use of IDS is | uired by Hospital Policy to utilize <u>Investigational Drug Service (IDS) pharmacies (Oncology</u> highly recommended, but optional for outpatient studies. Outpatient studies not using IDS c inspection by the IDS for compliance with drug accountability good clinical practices. |
| ndicate where study drug(s) w | vill be housed and managed: |
| Investigational Drug Ser | rvice (IDS) UK Hospital |
| Other Location: | |
| s the study being conducted u | under a valid Investigational New Drug (IND) application? |
| Yes ○ No | |
| If Yes, list IND #(s) and o | complete the following: |
| #69,214 | |
| J#09,214 | |
| IND Submitted/Hold by: | |
| IND Submitted/Held by: | |
| Sponsor: □ | Held By: |
| – | Held By: Sharon L. Walsh, PhD |
| Investigator: M | Tions 59. Sharon E. Walsh, Fild |
| Investigator: ਯ<br>Other: □ | Held By: |

For guidance and reporting requirements at the conclusion of treatment see the Expanded Access SOP.

Complete and attach the required <u>Study Drug Form</u> picking "Study Drug Form" for the document type. Any applicable drug documentation (e.g., Investigator Brochure; approved labeling; publication; FDA correspondence, etc.) should be attached using "Other Drug Documentation" for the document type.



# Attachments

| Attach Type | File Name |
|-----------------|------------------------------------|
| Study Drug Form | FDA IND Approval (19 May 2004).pdf |
| Study Drug Form | Form-o-Study-Drug-form.pdf |

#### STUDY DEVICE INFORMATION

0 unresolved comment(s)

Medical devices are intended for use in the diagnosis of disease or other conditions, or in the cure, mitigation, treatment, or prevention of disease, in man or other animals, or intended to affect the structure or any function of the body of man or other animals.

#### A DEVICE may be a:

- · component, part, accessory;
- assay, reagent, or in-vitro diagnostic device;
- software, digital health, or mobile medical app;
- other instrument if intended to affect the structure or function of the body, diagnose, cure, mitigate, treat or prevent disease; or
- a homemade device developed by an investigator or other non-commercial entity and not approved for marketing by FDA.

For additional information, helpful resources, and definitions, see ORI's <u>Use of Any Device Being Tested in Research web page</u>.

Does this protocol involve testing (collecting safety or efficacy data) of a medical device including an FDA approved device, unapproved use of an approved device, humanitarian use device, and/or an investigational device?

○ Yes ○ No

[Note: If a marketed device(s) is only being used to elicit or measure a physiologic response or clinical outcome, AND, NO data will be collected on or about the device itself, you may answer "no" above, save and exit this section, (Examples: a chemo drug study uses an MRI to measure tumor growth but does NOT assess how effective the MRI is at making the measurement; an exercise study uses a heart monitor to measure athletic performance but no safety or efficacy information will be collected about the device itself, nor will the data collected be used for comparative purposes against any other similar device).]

If you answered yes above, please complete the following questions.

| vice Name: | |
|---|---|
| he study being conducted | under a valid Investigational Device Exemption (IDE), |
| | ion (HDE) or Compassionate Use? |
| Yes No | |
| If Yes, complete the follo | owing: |
| IDE or HDE #(s) | |
| IDE/HDE Submitted/Hel | d by: |
| Sponsor: | Held By: |
| Investigator: □ | Held By: |
| Other: □ | Held By: |
| Check if this is a Tr<br>Expanded Access pro | eatment IDE or Compassionate Use under the Food and Drug Administration (FDA) |
| · | Group Expanded Access, see FDA's Early Expanded Access Program Information, |
| and attach the following | |
| | cess approval or sponsor's authorization; |
| | sessment from an uninvolved physician, if available;<br>reement from manufacturer or entity authorized to provide access to the product. |
| | reement from manufacturer or entity authorized to provide access to the product. |
| _ | ting requirements at the conclusion of treatment see the Medical Device SOP. |

Does the intended use of any research device being tested (not clinically observed) in this study meet the regulatory definition [FDA's PDF] of Significant Risk (SR) device?

∇es. Device(s) being tested in this study presents a potential for serious risk to the health, safety, or welfare of a subject and (1) is intended as an implant; or (2) is used in supporting or sustaining human life; or (3) is of substantial importance in diagnosing, curing, mitigating or treating disease, or otherwise prevents impairment of human health; or (4) otherwise presents a potential for serious risk to the health, safety, or welfare of a subject.

No. All devices being tested in this study do not present a potential for serious risk to the health, safety, or welfare of subjects/participants.

Complete and attach the required <u>Study Device Form</u>, picking the "Study Device Form" for the document type. Any applicable device documentation (e.g., Manufacturer information; patient information packet; approved labeling; FDA correspondence, etc.) should be attached using "Other Device Documentation" for the document type.



Attachments

RESEARCH SITES 0 unresolved comment(s)

To complete this section, ensure the responses are accurate then click "SAVE".

A) Check all the applicable sites listed below at which the research will be conducted. If none apply, you do not need to check any boxes.

#### **UK Sites**

- UK Classroom(s)/Lab(s)
- ☐ UK Clinics in Lexington
- □ UK Clinics outside of Lexington
- □ UK Healthcare Good Samaritan Hospital
- ∪K Hospital

#### Schools/Education Institutions

- □ Fayette Co. School Systems \*
- □ Other State/Regional School Systems
- ☐ Institutions of Higher Education (other than UK)

\*Fayette Co. School systems, as well as other non-UK sites, have additional requirements that must be addressed. See ORI's IRB Application Instructions - Off-site Research web page for details.

#### Other Medical Facilities

- □ Bluegrass Regional Mental Health Retardation Board
- □ Cardinal Hill Hospital
- □ Eastern State Hospital
- □ Norton Healthcare
- □ Nursing Homes
- □ Shriner's Children's Hospital
- □ Veterans Affairs Medical Center
- □ Other Hospitals and Med. Centers
- □ Correctional Facilities
- ☐ Home Health Agencies
- □ International Sites

Research activities conducted at performance sites that are not owned or operated by the University of Kentucky (UK) or at sites that do not fall under the UK IRB's authority, are subject to special procedures for coordination of research review. Additional information is required (see IRB Application Instructions - Off-Site Research web page), including:

- A letter of support and local context is required from non-UK sites. See *Letters of Support and Local Context* on the IRB Application Instructions Off-Site Research web page for more information.
- Supportive documentation, including letters of support, can be attached below. When attaching reliance documents, please ensure that you select the correct 'Document Type' from the drop-down menu. See below for the "Document Types" in bold, followed by examples of reliance documents for each type:
  - Individual Investigator Agreement (IIA)
    - A completed Individual Investigator Agreement

- IRB Approval (Non-UK)
  - A Letter of Approval from a Non-UK IRB
- IRB Authorization Agreement (IAA)
  - A SMART IRB Agreement
  - An OHRP Agreement
  - A DoD Agreement
  - An IREx Reliance Notification
  - Any Reliance Agreement
- Letter of Support & Local Context
  - A Letter of Support from an organization at which some research activities are occurring
  - Communications Plan
  - Local Context Form

Please reach out to <a href="mailto:IRBReliance@uky.edu">IRBReliance@uky.edu</a> if you have any questions or concerns.

- NOTE: If the non-UK sites or non-UK personnel are engaged in the research, there are additional federal and
  university requirements which need to be completed for their participation. For instance, the other site(s) may need
  to complete their own IRB review, or a cooperative review arrangement may need to be established with non-UK
  sites.
- Questions about the participation of non-UK sites/personnel should be discussed with the ORI staff at (859) 257-9428.

List all other non-UK owned/operated locations where the research will be conducted:

| UK Robert Straus Research Building | |
|---|---|
| Describe the role of any non-UK site(s) or nor | n-UK personnel who will be participating in your research. |
| Please describe the plan for the management protocol modifications and interim results from | t of reporting unanticipated problems, noncompliance, and submission of the non-UK sites: |
| Attachments | |

B) If your research involves collaboration with any sites and/or personnel outside the University of Kentucky, then it is considered multisite research and IRB reliance issues will need to be addressed. This may include national multi-center trials as well local studies involving sites/personnel external to UK. If you would like to request that the University of Kentucky IRB (UK IRB) serve as the lead IRB for your study, or if you would like the UK IRB to defer review to another IRB, please contact the <a href="mailto:IRBReliance@uky.edu">IRBReliance@uky.edu</a>.

#### RESEARCH ATTRIBUTES

0 unresolved comment(s)

Instructions: For various reasons, it is necessary to determine whether your research activities meet the definition of clinical research and/or a clinical trial. Your responses to the next series of questions will make that determination. For more details on the definitions, go to ORI's <u>clinical research vs. clinical trial web page</u> or visit <u>NIH's decision tree</u> for the NIH Clinical Trial definition.

Contact the Clinical Research Support Office (CRSO) if your study provides clinical services (e.g., labs, biopsies, tissue samples, physical exams, PT, counseling) regardless of payer (grant, federal, UK, industry)), utilizes UKHC space, or meets the NIH definition of a clinical trial (thereby requiring registry with CT.gov) as your study will need to be entered in OnCore to ensure appropriate regulatory tracking and billing. Visit <u>CRSO FAQs</u> for more information; requests for CCTS/CRSO services can be submitted via their <u>service request form</u>. For other questions, you can contact the CRSO Director, Jessica Heskel, at <a href="https://inhesk2@uky.edu">jhesk2@uky.edu</a>.

My research activities include one or more of the following:

Patient-oriented research regarding mechanisms of human disease, therapeutic interventions, clinical studies, or development of new technologies

Material of human origin (such as tissues, specimens, and cognitive phenomena) for which an investigator (or colleague) directly interacts with human subjects

Epidemiologic or Behavioral Studies

Outcomes Research or Health Services Research

Does your research study involve one or more human subjects prospectively assigned into one or more interventions (which may include placebo or other control) to evaluate the effects of those interventions on health-related biomedical or behavioral outcomes?

Indicate the items below that apply to your research. Depending on the items applicable to your research, you may be required to complete additional forms or meet additional requirements. Contact the ORI (859-257-9428) if you have questions about additional requirements.

□ Not applicable

-Check All That Apply-

- ☐ Academic Degree/Required Research
- ☑ Alcohol/Drug/Substance Abuse Research
- ☐ Biological Specimen Bank Creation (for sharing)
- ☐ Cancer Research
- □ Certificate of Confidentiality
- □ Collection of Biological Specimens for banking and use
- □ Community-Based Participatory Research
- □ Deception
- □ Educational/Student Records (e.g., GPA, test scores)
- □ Emergency Use (Single Patient)
- ☐ Gene Transfer

For additional requirements and information:

- Cancer Research (MCC PRMC)
- <u>Certificate of Confidentiality</u> (look up "Confidentiality/Privacy...")
- CCTS (Contex for Clinical a
- CCTS (Center for Clinical and Translational Science)
- <u>Clinical Research</u> (look up "What is the definition of....)
- Clinical Trial
- Collection of Biological Specimens for Banking (look up "Banks, Repositories, Registries...")
- <u>Collection of Biological Specimens</u> (look up "Repositories, Registries, Specimen/Tissue Banks...")
- <u>Community-Based Participatory Research</u> (look up "Community-Engaged...")
- Data & Safety Monitoring Board (DSMB)

\*For Medical IRB: <u>Service Request Form</u> for CCTS DSMB

- Data & Safety Monitoring Plan
- Deception\*

- ☐ Genetic Research
- □NIH Genomic Data Sharing (GDS) (databases such as GWAS, dbGaP, GenBank)
- $\hfill\Box$  Treatment with Human Cells, Tissues, and Cellular and Tissue Based Products
- □ Individual Expanded Access or Compassionate Use
- □ International Research
- □ Planned Emergency Research Involving Exception from Informed Consent
- □ Recombinant DNA
- □ Registry or data repository creation
- □ Stem Cell Research
- □ Suicide Ideation or Behavior Research
- □ Survey Research
- □ Transplants
- $\hfill\square$  Use, storage and disposal of radioactive material and radiation producing devices
- □ Vaccine Trials

- \*For deception research, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"
- Emergency Use (Single Patient) [attach Emergency Use Checklist] (PDF)
- Genetic Research (look up "Banks, Repositories, ...Genetic/Genomic Data Sharing...")
- Gene Transfer

\*For gene transfer research, also go to the E-IRB Application Other Review Committees section, and checkmark Institutional Biosafety Committee

- International Research (look up "International & Non-English Speaking")
- NIH Genomic Data Sharing (GDS) Policy (PDF)
- Planned Emergency Research Involving Exception to Informed Consent\*

\*For Planned Emergency Research Involving Waiver of Informed Consent, also go to the E-IRB Application Informed Consent section, checkmark and complete "Request for Waiver of Informed Consent Process"

 Use, storage and disposal of radioactive material and radiation producing devices

# FUNDING/SUPPORT 0 unresolved comment(s)

If the research is being submitted to, supported by, or conducted in cooperation with an external or internal agency or funding program, indicate below all the categories that apply. •

□ Not applicable

#### -Check All That Apply-

☐ Grant application pending

☑ (NIH) National Institutes of Health

□(CDC) Centers for Disease Control & Prevention

☐ (HRSA) Health Resources and Services

Administration

☐ (SAMHSA) Substance Abuse and Mental Health Services Administration

□(DoJ) Department of Justice or Bureau of Prisons

□ (DoE) Department of Energy

□ (EPA) Environmental Protection Agency

□ Federal Agencies Other Than Those Listed Here

□ Industry (Other than Pharmaceutical Companies)

□ Internal Grant Program w/ proposal

□ Internal Grant Program w/o proposal

□ National Science Foundation

☐ Other Institutions of Higher Education

□ Pharmaceutical Company

□ Private Foundation/Association

□ U.S. Department of Education

□ State

Other:

Click applicable listing(s) for additional requirements and information:

- (HHS) Dept. of Health & Human Services
- (NIH) National Institutes of Health
- (CDC) Centers for Disease Control & Prevention
- (HRSA) Health Resources & Services Administration
- (SAMHSA) Substance Abuse & Mental Health Services Administration
- Industry (Other than Pharmaceutical Companies) [IRB Fee Info-look up "Does the IRB Charge a Fee..."]
- National Science Foundation
- (DoEd) U.S. Department of Education
- (DoJ) Department of Justice or Bureau of Prisons
- (DoE) Department of Energy Summary and Department of Energy Identifiable Information Compliance Checklist
- (EPA) Environmental Protection Agency

Specify the funding source and/or cooperating organization(s) (e.g., National Cancer Institute, Ford Foundation, Eli Lilly & Company, South Western Oncology Group, Bureau of Prisons, etc.):

National Institute on Drug Abuse

#### Add Related Grants

If applicable, please search for and select the OSPA Account number or Electronic Internal Approval Form (eIAF) # (notif #) associated with this IRB application using the "Add Related Grants" button.

If required by your funding agency, upload your grant using the "Grant/Contract Attachments" button.

Add Related Grants

**Grant/Contract Attachments** 

| Attach Type | File Name |
|---------------|--------------------|
| GrantContract | Grant Proposal.pdf |

The research involves use of Department of Defense (DoD) funding, military personnel, DoD facilities, or other DoD resources. (See <u>DoD SOP</u> and <u>DoD Summary</u> for details)

Using the "attachments" button (below), attach applicable materials addressing the specific processes described in the DoD SOP.

Additional Certification: (If your project is federally funded, your funding agency may request an Assurance/ Certification/Declaration of Exemption form.) Check the following if needed:

□ Protection of Human Subjects Assurance/Certification/Declaration of Exemption (Formerly Optional Form – 310)

Assurance/Certification Attachments

#### OTHER REVIEW COMMITTEES

0 unresolved comment(s)

If you check any of the below committees, additional materials may be required with your application submission.

Does your research fall under the purview of any of the other review committees listed below? [If yes, check all that apply and attach applicable materials using the attachment button at the bottom of your screen.]

∩ Yes ∩ No

#### □ Institutional Biosafety Committee

- □ Radiation Safety Committee
- □ Radioactive Drug Research Committee
- ☐ Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC)
- ☐ Graduate Medical Education Committee (GME)
- ☐ Office of Medical Education (OME)

#### **Additional Information**

- Institutional Biosafety Committee (IBC) Attach required IBC materials
- Radiation Safety Committee (RSC) For applicability, see instructions
- Radioactive Drug Research Committee (RDRC)
- Markey Cancer Center (MCC) Protocol Review and Monitoring <u>Committee (PRMC)\*\*</u> - Attach MCC PRMC materials, if any, per instructions.
- Office of Medical Education (OME)
- Graduate Medical Education Committee (GME)

### Attachments

\*\* If your study involves cancer research, be sure to select "Cancer Research" in the "Research Attributes" section. ORI will send your research protocol to the Markey Cancer Center (MCC) Protocol Review and Monitoring Committee (PRMC). The MCC PRMC is responsible for determining whether the study meets the National Cancer Institute (NCI) definition of a clinical trial and for issuing documentation to you (the investigator) which confirms either that PRMC approval has been obtained or that PRMC review is not required. Your IRB application will be processed and reviewed independently from the PRMC review.

#### ADDITIONAL INFORMATION/MATERIALS

0 unresolved comment(s)

Do you want specific information inserted into your approval letter? OYes ONo

Approval Letter Details:

If you wish to have specific language included in your approval letter (e.g., serial #, internal tracking identifier, etc...), type that language in the box below exactly as it should appear in the letter. The text you enter will automatically appear at the top of all approval letters, identical to how you typed it, until you update it. Don't include instructions or questions to ORI staff as those will appear in your approval letter. If these details need to be changed for any reason, you are responsible for updating the content of this field.

| Additional | Materials: |
|------------|------------|

If you have other materials you would like to include for the IRB's consideration, check all that apply and attach the corresponding documents using the Attachments button below.

□ Detailed protocol

□ Dept. of Health & Human Services (DHHS) approved protocol (such as NIH sponsored Cooperative Group Clinical Trial)

Other Documents

Protocol/Other Attachments

#### Attach Type File Name

Other Progress Report - Opioids & Alcohol - 08.18.2025.pdf

NOTE: Instructions for Dept. of Health & Human Services (DHHS)-approved protocol

If you have password protected documents, that feature should be disabled prior to uploading to ensure access for IRB review.

To view the materials currently attached to your application, click "All Attachments" on the left menu bar.

#### SIGNATURES (ASSURANCES)

0 unresolved comment(s)

#### Introduction

All IRB applications require additional assurances by a Department Chairperson or equivalent (DA), and when applicable, a Faculty Advisor or equivalent (FA). This signifies the acceptance of certain responsibilities and that the science is meritorious and deserving of conduct in humans. The person assigned as DA should not also be listed in the Study Personnel section, and the individual assigned as FA should be listed in the Study Personnel section.

For a list of responsibilities reflected by signing the Assurance Statement, refer to "What does the Department Chairperson's Assurance Statement on the IRB application mean?"

For a detailed illustration of how to complete this section, please review the short online video tutorial <u>"Signatures (Assurance) Section - How to Complete,"</u> Otherwise, follow the steps below.

### **Required Signatures:**

Individuals chosen as signees may remove the application from their Inbox without signing the Assurance Statement by clicking "Return to PI" with a comment about why it is being returned (e.g., specific edits are deemed necessary).

The PI, and personnel chosen as a contact, will receive an email notification that edits are needed, and can find the draft application in both the "Draft" folder and the "Signatures Status" folder located in the menu in the left margin of the default Inbox page. The researcher does not have a 'reply' option to the signee's comments and must make the requested edits directly in the application, or communicate outside the E-IRB system as to why not. Once the response is finalized, the researcher must re-visit the "Assurances Required" section to click the "Return to Signee" button for their reconsideration; the signee will receive an email notification at that time.

Hover your mouse cursor here for additional instructions.

| 0 | | | | | | |
|---|---|---|---|---|---|---|
| First<br>Name | Last<br>Name | Role | Department | Signee<br>Return<br>Comment | Date<br>Signed | |
| Thomas | Kelly | Department<br>Authorization | Behavioral<br>Science | | 11/19/2019<br>03:40 PM | View/Sign |
| Sharon | Walsh | Principal<br>Investigator | Behavioral<br>Science | | 11/19/2019<br>10:24 AM | View/Sign |

#### **Department Authorization**

™ This is to certify that I have reviewed this research protocol and that I attest to the scientific validity and importance of this study; to the qualifications of the investigator(s) to conduct the project and their time available for the project; that facilities, equipment, and personnel are adequate to conduct the research; and that continued guidance will be provided as appropriate. When the principal investigator assumes a sponsor function, the investigator has been notified of the additional regulatory requirements of the sponsor and by signing the principal investigator Assurance Statement, confirms he/she can comply with them.

\*If the Principal Investigator is also the Chairperson of the department, the Vice Chairperson or equivalent should complete the "Department Authorization".

\*\*IF APPLICABLE FOR RELIANCE: I attest that the principal investigator has been notified of the regulatory requirements of both the Reviewing and Relying IRBs, according to the information provided in the E-IRB application. The attached Reliance Assurance Statement, signed by the principal investigator, confirms that he/she can comply with both sets of IRB requirements.

I understand the University of Kentucky's policies concerning research involving human subjects and I agree:

- 1. To comply with all IRB policies, decisions, conditions, and requirements;
- 2. To accept responsibility for the scientific and ethical conduct of this research study;
- 3. To obtain prior approval from the Institutional Review Board before amending or altering the research protocol or implementing changes in the approved consent/assent form;
- 4. To report to the IRB in accord with IRB/IBC policy, any adverse event(s) and/or unanticipated problem(s) involving risks to subjects;
- 5. To complete, on request by the IRB for Full and Expedited studies, the Continuation/Final Review Forms;
- To notify the Office of Sponsored Projects Administration (OSPA) and/or the IRB (when applicable) of the development of any financial interest not already disclosed;
- 7. Each individual listed as study personnel in this application has received the mandatory human research protections education (e.g., CITI);
- 8. Each individual listed as study personnel in this application possesses the necessary experience for conducting research activities in the role described for this research study.
- 9. To recognize and accept additional regulatory responsibilities if serving as both a sponsor and investigator for FDA regulated research.

**☑** Furthermore, by checking this box, I also attest that:

- I have appropriate facilities and resources for conducting the study;
- I am aware of and take full responsibility for the accuracy of all materials submitted to the IRB for review;
- If applying for an exemption, I also certify that the only involvement of human subjects in this research study will be in the categories specified in the Protocol Type: Exemption Categories section.
- If applying for an Abbreviated Application (AA) to rely on an external IRB, I understand that certain items above (1, 3, 4, 7-8) may not apply, or may be altered due to external institutional/IRB policies. I document my agreement with the <a href="Principal Investigator Reliance Assurance Statement">Principal Investigator Reliance Assurance Statement</a> by digitally signing this application.

\*You will be able to "sign" your assurance after you have sent your application for signatures (use Submission section). Once all Assurance Statement signatures have been acquired, return to this section to submit your application to ORI.

#### SUBMISSION INFORMATION

0 unresolved comment(s)

\*\*\* If this Continuation Review entails a change in the scope of your activities to include COVID-19 related research, please insert "COVID19" at the start of your Project and Short Titles.\*\*\*

Each Section/Subsection in the menu on the left must have a checkmark beside it (except this Submission section) indicating the Section/Subsection has been completed. Otherwise your submission for IRB review and approval cannot be sent to the Office of Research Integrity/IRB.

If applicable, remember to update the Approval Letter Details text box under the Additional Information section

If your materials require review at a convened IRB meeting which you will be asked to attend, it will be scheduled on the next available agenda and you will receive a message to notify you of the date.

If you are making a change to an attachment, you need to delete the attachment, upload a highlighted version that contains the changes (use Document Type of "Highlighted Changes"), and a version that contains the changes without any highlights (use the appropriate Document Type for the item(s)). Do **not** delete approved attachments that are still in use.

Principal Investigator's Assurance Statement

I understand the University of Kentucky's policies concerning research involving human subjects, and I attest to:

- 1. Having reviewed all the investigational data from this study, including a compilation of all internal and external unanticipated problems.
- 2. Having reviewed, if applicable, information from the sponsor including updated investigator brochures and data and safety monitoring board reports.

I also attest that I have reviewed pertinent materials concerning the research and concluded either:

- A. The human subject risk/benefit relationship is NOT altered, and that it is not necessary to modify the protocol or the informed consent process,
   OR.
- B. The human subject risk/benefit relationship has been altered, and have previously submitted or am including with this continuation review submission, a modification of the research protocol and informed consent process.

■ By checking this box, I am providing assurances for the applicable items listed above.

Your protocol has been submitted.

# Download all

| | Document Type | File Loaded | Document Description | File<br>Size | Modified<br>By | Mod Date |
|---|---|---|---|---|---|---|
| 4 | ApprovalLetter | ApprovalLetter.pdf | | 0.090 | jchine2 | 9/2/2025<br>9:32:09 AM |
| 4 | AddInfoProduct | Progress Report - Opioids &<br>Alcohol - 08.18.2025.pdf | Progress Report dated 18AUG2025 | 0.111 | mmdo225 | 8/20/2025<br>1:23:16 PM |
| 4 | CR_EntireConsent | Signed Consents - 1 Screening & 1 Main Study.pdf | Signed Consents - 1 Screening & 1 Main Study | 1.148 | mmdo225 | 8/18/2025<br>11:42:15<br>AM |
| 4 | StudyDesign | Opioids & Alcohol Pilot Phase<br>Completion 2-14-2023.docx | Pilot phase completion | 0.013 | sbr333 | 2/14/2023<br>2:05:40 PM |
| 4 | Advertising | Opioids & Alcohol Digital Ads 6.8.22 (CLEAN).pdf | Opioids & Alcohol Digital Ads, 6.8.22, Clean Copy | 0.993 | sbr333 | 6/14/2022<br>10:43:14<br>AM |
| 4 | Advertising | Opioid & Alcohol - Digital ads<br>6.8.22 (PR APPROVED).pdf | Opioids & Alcohol Digital Ads, 6.8.22, PR Stamped | 1.947 | sbr333 | 6/14/2022<br>10:42:28<br>AM |
| 4 | Advertising | Opioid & Alcohol Flyers 6.8.22 (PR APPROVED).pdf | Opioids & Alcohol Flyers, 6.8.22, PR<br>Stamped | 3.832 | sbr333 | 6/14/2022<br>10:42:00<br>AM |
| 4 | Advertising | Opioid & Alcohol - Cards 6.8.22<br>(PR Approved).pdf | Opioids & Alcohol Card Ads, 6.8.22,<br>PR Stamped | 5.854 | sbr333 | 6/14/2022<br>10:41:29<br>AM |
| 4 | Advertising | Opioid & Alcohol - Cards 6.8.22<br>(CLEAN).pdf | Opioid & Alcohol card ads, 6.8.22,<br>Clean Copy | 5.799 | sbr333 | 6/14/2022<br>10:32:28<br>AM |
| 4 | Advertising | Opioid & Alcohol Flyer 6.8.22<br>(CLEAN).pdf | Opioid & Alcohol Flyers, 6.8.22,<br>Clean Copy | 3.799 | sbr333 | 6/14/2022<br>10:31:27<br>AM |
| 4 | Advertising | Tracked Changes - BuildClinical<br>Secure questionnaire.pdf | Tracked Changes - BuildClinical<br>Secure Questionnaire | 0.083 | mmdo225 | 3/2/2022<br>11:10:02<br>AM |
| 4 | Advertising | BuildClinical Secure questionnaire.pdf | BuildClinical Secure questionnaire | 0.039 | mmdo225 | 2/8/2022<br>12:53:43<br>PM |
| 4 | Advertising | BuildClinical Opioid ads - PR stamped.pdf | BuildClinical Opioid ads - PR stamped | 0.718 | mmdo225 | 2/8/2022<br>12:53:25<br>PM |
| 4 | Advertising | BuildClinical Landing Page - PR stamped.pdf | BuildClinical Landing Page - PR stamped | 1.174 | mmdo225 | 2/8/2022<br>12:53:05<br>PM |
| 4 | AdditionInfoConsiderations | Progress Report - Opioids<br>Alcohol.pdf | Progress Report - Opioids Alcohol | 0.070 | sbr333 | 10/5/2021<br>12:18:46<br>PM |
| 4 | Advertising | Possible Accompanying Text for Online Ads APPROVED.pdf | Opioids & Alcohol PR Approved Online Ad Accompanying Text | 0.148 | sbr333 | 3/25/2020<br>11:18:18<br>AM |
| 4 | Advertising | Opioid & Alcohol ads (clean).pdf | Opioid & Alcohol Ads, Clean Copy | 18.444 | sbr333 | 3/25/2020<br>11:14:22<br>AM |
| 4 | DataCollection | Session Questionnaires - 03.20.2020.pdf | Opioid & Alcohol Session<br>Questionnaires | 0.175 | mmdo225 | 3/23/2020 |
| 4 | DataCollection | Screening Questionnaires - 03.20.2020.pdf | Opioid & Alcohol Screening Questionnaires | 1.092 | mmdo225 | 3/23/2020 |
| 4 | Advertising | 20201 Op x alcohol PR approved ads - 03.20.2020.pdf | Opioid & Alcohol PR Approved Ads | 17.289 | mmdo225 | 3/23/2020<br>3:14:51 PM |
| 4 | StudyDrug | Form-o-Study-Drug-form.pdf | Study Drug Form | 0.438 | sbr333 | 11/13/2019<br>11:33:30<br>AM |
| 4 | StudyDrug | FDA IND Approval (19 May 2004).pdf | | 0.060 | sbr333 | 11/6/2019<br>11:18:04<br>AM |

| | | | | | | 55176 |
|---|---|---|---|---|---|---|
| 4 | Advertising | Facebook page - revised Dec 17<br>APPROVED.pdf | Facebook Page | 0.626 | sbr333 | 10/24/2019<br>11:54:04<br>AM |
| 4 | GrantContract | Grant Proposal.pdf | Grant Proposal | 1.218 | sbr333 | 10/24/2019<br>11:50:42<br>AM |

Protocol Number: 55176

### Protocol Changes

Click link to sort Changed Date Expedited Categories XPCategory0 changed by mmdo225 on 8/26/2025 9:30:15 AM

Y
Expedited Categories XPCategory1 changed by mmdo225 on 8/26/2025 9:30:15 AM
Expedited Categories XPCategory2 changed by mmdo225 on 8/26/2025 9:30:15 AM

Expedited Categories XPCategory3 changed by mmdo225 on 8/26/2025 9:30:15 AM Expedited Categories XPCategory4 changed by mmdo225 on 8/26/2025 9:30:15 AM Expedited Categories XPCategory4 changed by mmdo225 on 8/26/2025 9:30:15 AM

N Expedited Categories XPCategory5 changed by mmdo225 on 8/26/2025 9:30:15 AM

N Expedited Categories XPCategory6 changed by mmdo225 on 8/26/2025 9:30:15 AM

N
Expedited Categories XPCategory7 changed by mmdo225 on 8/28/2025 9:30:15 AM
N
Informed Consent InformedConsentHPAACombinedForm changed by mmdo225 on 8/18/2025 11:59:28 AM

Informed Consent InformedConsentHPAACombinedForm changed by mindo225 on 8 No Informed Consent StampedConsent changed by mindo225 on 8 /18/2025 11.59:28 AM NO Information ProjectEndDate changed by mindo225 on 8 /18/2025 11.57:41 AM 6/30/20262 12:00:00 AM Project Information SubjectCount changed by mindo225 on 8 /18/2025 11.57:56 AM 72/4 Risk Level RiskCategory changed by mindo225 on 8 /18/2025 11.58:44 AM 31 Study Personnel Changes:

| Status | PPIdentity | ProtocoIID | PersonID | RoleInProtocol | IsContact | LastNam | e FirstNam | e Email | DeptCode | RoomBuilding | SpeedSort | PhoneNum | DeptDesc | AuthorizedConsent | ResponsibilityInProject | Degree | Rank | StatusFlag | IsRemoved | ModBy ModDate | SFI IsPIRN MiddleNam |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Deleted | 1088665 | 107174 | 12374202 | SP | N | Oller | Devin | Devin.Oller@uky.edu | | | | | | N | Consultant/Advisor | | | | Υ | mmdo225 8/20/2025<br>11:29:36<br>AM | N |
| Deleted | 1088681 | 107174 | 12599499 | SP | N | McGee | Paul | pwmc226@uky.edu | | | | | | Υ | Data Collection | | | Р | Υ | mmdo225 8/20/2025<br>1:37:30<br>PM | N |

55176

### Protocol Type Comment by Lindsay Schneider - ORI to IRB/PI on 8/25/2025 3:14:09 PM

Based on your answer to Question #1 in the Continuation Review (CR) Form, this protocol now qualifies for Expedited Review. Your CR request has been returned so that you can make the following changes:

- 1. Revise the PROTOCOL TYPE section to be Expedited.
- 2. Checkmark the EXPEDITED CATEGORY "originally approved by Full IRB at convened meeting".
- 3. Re-submit the revised protocol.

Be sure to complete these tasks with enough leeway for Expedited Review before approval lapse on 10/07/2025.

When you re-submit, your protocol will be managed by Joanne Hines, who manages the MEDXP Dashboard for IRB #2.

If you feel you received this message in error, please revisit your CR Form and then contact Lindsay Schneider at Irsc222@uky.edu or 859-562-0647. Thank you!

Interactions of Alcohol and Opioids: Pharmacodynamic Effects

Protocol Number 55176

NCT: 04300751

# **Statistical Analysis Plan for Primary Study**

#### 1. Introduction

The purpose of this document is to provide details about the study population, how missing data will be handled, and the statistical methodologies that will be used to analyze the data for the primary study.

### 2. General Conventions

All analyses will be conducted using SAS Version 9.3 or higher (SAS Institute, Inc; Cary, NC, USA), and all hypothesis testing will be two-sided with a significance level of 0.05. P-values will be presented with 3 decimals and p-values that are less than 0.001 will be represented as <0.001.

Continuous data will be summarized using descriptive statistics: number of observations (n), arithmetic mean, standard error, minimum, and maximum. Frequencies and percentages will be used to summarize categorical (discrete) outcomes. Means and standard errors will be presented to two decimal places.

### 3. Analysis Populations

Two study populations will be defined for analysis.

# 3.1 Enrolled Population

All subjects who sign the Informed Consent Form.

# 3.2 Completer Population

Subjects in the who complete the entire Study Phase.

# 4. Subjects and Demographics

# 4.1 Disposition and Withdrawals

Subject disposition will be summarized using the number and percent of subjects who are in the Enrolled Population and Completer Population.

# 4.2 Demographics and Other Baseline Characteristics

Demographic and baseline characteristics will be summarized for the Completer Population. No statistical comparisons will be made on demographic or baseline

characteristics. The demographic and baseline characteristics will consist of age, sex, race, ethnicity, height (cm), weight (kg), and BMI (kg/m²).

Continuous variables (age, height, weight, BMI) will be summarized by n, mean, standard deviation, min, median, and max. Frequencies and percentages will be used to describe categorical (discrete) variables including gender, race, and ethnicity.

# 5. Pharmacodynamic Analyses

# 5.1 Primary Pharmacodynamic Analyses

The primary analyses will be performed based on the Completer Population. The primary Emax VAS item Drug Liking and will be analyzed in a mixed model including the nine drug conditions with a compound symmetry covariance structure. Within each model, subject will be treated as random effects, and the remaining parameter as fixed effects. Mixed models are suited for data with repeated measures, correlations among observations within an individual subject, and the presence of missing data. The response of individual subjects is first modeled, and then the estimates for each individual are combined in a group analysis (Singer, 1998; Ballinger 2004; Diggle et al. 1996; Gibbons et al. 1993; Kreft and De Leeuw 1998). Tukey post-hoc tests will compare active doses to placebo and other relevant active dose comparisons.

# **5.2 Secondary Pharmacodynamic Analyses**

Secondary analyses will be performed based on the Completer Population. Secondary pharmacodynamic outcomes will include:

- Raw time course data of VAS items (e.g., High, Good Drug Effects, Bad Drug Effects, Any Drug Effects, Desire to Use Opioids), subjective opioid adjectives, street value, observer adjectives, DSST, cold pressor test, cold water VAS, flicker/fusion, balance task, heart rate, systolic blood pressure, diastolic blood pressure, respiration rate, oxygen saturation, end tidal carbon dioxide, and pupil diameter from the nine dose conditions.
- Emax and Emin (where appropriate) on the VAS items, subjective opioid adjectives, street value, observer adjectives, DSST, cold pressor test, cold water VAS, flicker/fusion, balance task, heart rate, systolic blood pressure, diastolic blood pressure, respiration rate, oxygen saturation, end tidal carbon dioxide, and pupil diameter from the nine dose conditions.

Secondary analyses will be completed in mixed models that include drug condition and time (when appropriate with an autoregressive covariance structure) with a compound symmetry covariance structure. Subject will be treated as random effects and the remaining parameters fixed. Tukey post-hoc tests will compare active doses to placebo and other relevant active dose comparisons.

**5.2.1 Drug Identification Assessments:** Drug identification assessments completed during the experimental dose sessions will be summarized by frequencies and percentages to describe categorical outcomes.

# 6. Safety and Tolerability Analyses

Safety analyses will be performed on the Enrolled Population. Adverse events (AEs) recorded after signing informed consent but prior to the first dose will be recorded as baseline AEs and will be listed by subject but will not be included in the summary safety analysis. AEs will be summarized by relationship to study drug and severity.

The numbers and frequencies of subjects reporting AEs, including abuse-related AEs, will be summarized. If the same AE (preferred term) is reported more than once for the same subject, it will only appear once in the summary tables and the highest severity grade and strongest relationship to treatment will be included in the summary. Any AEs leading to a study discontinuation will be summarized.

All deaths, other SAEs, and AEs will be listed.

Other safety variables, including clinically significant changes in the participant's physical examination, vital signs, electrocardiograms, and clinical laboratory results, will be tabulated and presented by study drug received.

# 7. Missing Data

Within-session missing data are expected to be less than 3% for each outcome. Inspection of missing data and correlates of missingness will be examined upon study completion. The use of mixed models as an analytic strategy obviates the need for the missing values to be imputed.

## 8. Identification and Summary of Protocol Deviations

Major protocol deviations from the participant's entry criteria through study completion will be documented and summarized as far as they can be extracted from the numeric and coded study data.

### References:

Ballinger GA (2004) Using generalized estimating equations for longitudinal data analysis. Organizational Research Methods 7(2): 127-150.

Diggle PJ, Liang K, Zeger SL (1996) Analysis of Longitudinal Data. Oxford University Press, Inc., Oxford University Press, Inc.

Gibbons RD, Hedeker D, Elkin I, Waternaux C, Kraemer HC, Greenhouse JB, Shea MT, Imber SD, Sotsky SM, Watkins JT (1993) Some conceptual and statistical issues in

analysis of longitudinal psychiatric data. Application to the NIMH treatment of Depression Collaborative Research Program dataset. Arch Gen Psychiatry 50: 739-50.

Kreft I, De Leeuw J (1998) Introducing Multilevel Modeling. Sage Publications, Ltd., Sage Publications, Ltd.

Singer JD (1998) Using SAS PROC MIXED to fit multilevel models, hierarchical models, and individual growth models. J Educ Behav Stat 24: 323-355.



### Consent and Authorization to Participate in a Research Study

#### **KEY INFORMATION FOR**

#### **MAIN STUDY CONSENT:**

#### THE BEHAVIORAL EFFECTS OF OPIOIDS AND ALCOHOL

You are being invited to take part in a research study about the effects of alcohol and opioid (examples: oxycodone, tramadol, codeine, hydrocodone) medications when taken alone and in combination. We plan to screen approximately 75 participants and plan to have up to 18 complete the study. This page is to give you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

By doing this study, we hope to learn about the effects of opioids and alcohol, and their effects on mood and behavior. Your participation in this research will include an approximately 30-night stay at the UK hospital (you will not be allowed to leave or have visitors during this time) and a short (about 3 hours) follow-up appointment approximately 2 weeks after leaving the hospital.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

There is no direct benefit to you for taking part in this study. Your willingness to participate may help us understand how alcohol and opioids affect your body, mood, and behavior. For a complete description of benefits, refer to Detailed Consent.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

If you are not between the ages of 21 and 55, if you have any serious medical condition(s) (for example, diabetes) or if you experience withdrawal when not using opioid drugs or alcohol, you should not participate in this study. If you are pregnant, planning on becoming pregnant, or nursing, you should not participate. If you are seeking treatment for substance use, you should not participate, and we will help you find treatment. You may choose not to participate if you are not able to live at the UK hospital for about a month. Let us know if that is a concern for you. There are also risks related to the use of study medications—a complete description of risks, including a full list of study medication side effects, are listed in the detailed portion of the consent form.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights you would normally have if you choose not to volunteer.

#### WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS OR CONCERNS?

If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study contact Sharon L. Walsh, Ph.D. of the University of Kentucky, Department of Behavioral Science and Center on Drug and Alcohol Research at (859) 257-6485.

If you have any concerns or questions about your rights as a volunteer in this research, contact staff in the University of Kentucky (UK) Office of Research Integrity (ORI) between the business hours of 8am and 5pm EST, Monday-Friday at 859-257-9428 or toll free at 1-866-400-9428.

#### **DETAILED CONSENT:**

#### ARE THERE REASONS WHY YOU WOULD NOT QUALIFY FOR THIS STUDY?

You will not be allowed to participate in the study if you are: under 21 or over 55 years of age; pregnant, breastfeeding, or planning on becoming pregnant; seeking treatment for your substance use; you do not use opioids for non-medical purposes (to get high, feel relaxed), or do not drink alcohol. You will not be allowed to participate if you are physically dependent on opioids, benzodiazepine/sedative-like drugs, or alcohol; however, we will provide treatment referrals to you if you are seeking treatment for your drug/alcohol use. You will not be allowed to participate if the medical staff thinks that giving you the study drugs could be dangerous to your health. If you have any serious medical problems (e.g., a history of heart problems, breathing problems, head trauma, epilepsy, or seizures), you will not be allowed to participate in this study. If you decide that you do not want to participate or do not think the study will fit your schedule, you should not take part.

#### WHERE WILL THE STUDY TAKE PLACE AND WHAT IS THE TOTAL AMOUNT OF TIME INVOLVED?

If you are selected to participate, you will live at the UK hospital Center for Clinical and Translational Science (CCTS) Clinical Research Unit (CRU). During your stay you will participate in 10 sessions. Each session will last approximately 7 hours and you will typically participate in 2 or 3 sessions per week. You will live on the inpatient unit for approximately 1 month and participate in sessions for about 70 hours across the whole month. You will be given a calendar that will list the date of each session. On your days off from session, you can read, watch movies, and engage in recreational activities, but you will not be permitted to leave the hospital or have visitors.

#### WHAT WILL YOU BE ASKED TO DO?

If you agree to participate in the study, we will ask you to do the following things:

- 1. Once you are medically cleared for the study, you will be admitted to the CCTS-CRU at the UK hospital. You may be asked to share a room with another volunteer of the same gender.
- 2. You will need to follow the inpatient unit rules while you are in the study. If you do not follow the rules, you will be removed from the study you will not receive a payment bonus if you are discharged for breaking rules. Some examples of these rules are:
  - You will not be allowed to have any visitors, but you will be able to make phone calls
  - You will be allowed to smoke cigarettes, but only under supervision of the CRU nursing staff in the outdoor designated smoking area
  - No sexual behavior or sexual intercourse for the duration of the study
  - No drug or alcohol use; you cannot use any drugs that are not given to you as part of the study
- 3. After you are admitted to the inpatient unit, we will show you the session room where testing will take place. We will teach you how to use the computer and show you the kinds of questions you will be asked and tasks you will need to complete. You will have plenty of time to ask questions about how to perform any of the tasks.
- 4. There will be a total of 10 sessions. The first session is a qualification session this session will help us determine if you will qualify for the rest of the study. If you continue to qualify, you will complete 9 experimental sessions. You will receive a calendar with the actual dates of your sessions, but a sample calendar with session dates is provided below. A more detailed calendar can be found in the Appendix section at the end of this packet.

#### Sample Study Calendar:

| | Sunday | Monday | Tuesday | Wednesday | Thursday | Friday | Saturday |
|---|---|---|---|---|---|---|---|
| Week 1 | | Admission | Practice/<br>Training | Session 1 -<br>Qualification | | Session 2 | |
| Week 2 | | Session 3 | | Session 4 | | Session 5 | |
| Week 3 | | Session 6 | | Session 7 | | Session 8 | |
| Week 4 | | Session 9 | | Session 10 | Discharge | | |

- 5. The first session is a qualification session to help us determine if you will qualify for the rest of the study. During the qualification session, you will receive a capsule to swallow– this capsule will contain either an opioid drug, (for example: hydromorphone, oxycodone, morphine, or hydrocodone) or placebo (an inactive substance). After you complete this session, you will be informed whether you qualify to continue with the rest of the study. If you do not qualify, you will be discharged. If you qualify, you will complete 9 additional experimental sessions.
- 6. During each of the 9 sessions, you will be asked to take capsules that contain a dose of an opioid drug (such as oxycodone, tramadol, codeine, hydrocodone). You will also be asked to drink a cocktail with or without an active dose of alcohol. Neither you nor the research staff will know what drug or alcohol dose you will receive on any particular day.
- 7. During sessions, we will measure how you respond to each of the doses by recording things like heart rate, blood pressure, oxygen saturation, expired carbon dioxide, respiration rate, and pupil diameter. We will also ask you questions about how you are feeling. For example, we may ask you if you like the drug effects or if you are feeling sick. We will also ask you to complete tasks that measure your coordination and balance and look at blinking lights to test your eyes this test will not harm your vision.

You will also participate in a cold-water task during each session. We will ask you to place your arm into a cooler of cold water and tell us when you start to feel pain and when you no longer wish to tolerate it. When you can no longer tolerate the cold water, you can remove your arm from the cooler. This task will not cause any lasting harm, and the pain will subside within a few minutes. We will ask you several questions about the pain you experienced during the task.

During session, you may engage in activities such as reading, as long as these activities do not interfere with the study or any of the scheduled tasks or questionnaires.

- 8. On days when you are not in session, you will be asked to fill out questionnaires each day. For example, we will ask you about how you feel, whether you feel tired or have an upset stomach. The nurses will measure your vital signs (heart rate, blood pressure, etc.) several times every day. You will also give breath and urine samples every day, which will be tested for drugs and alcohol; women will be tested for pregnancy.
- 9. If you are female, you will be tested regularly to see if you are pregnant. If the test is positive, you will be notified, discharged from the study, and referred for treatment. If you become pregnant at any time during the study (during screening, while you are in the hospital, in the time between study discharge and your follow-up appointment, or anytime in the 30 days after you leave the study), you will need to notify the study investigator (Sharon Walsh, Ph.D (859) 257-6485) or the study physician (Michelle Lofwall, M.D. (859) 323-9321).

By signing this consent form you are agreeing to practice an effective method of birth control (e.g., oral contraceptives, intrauterine device, diaphragm, condom) for the entire study duration (prior to study admission through 30 days after study completion).

- 10. After you have completed all sessions, you will be discharged from the study. We will ask you to complete a follow-up appointment approximately 2 weeks after discharge. We will ask you about your health and drug use. You will be paid \$25. The follow-up appointment may be conducted over the phone or in person at the Robert Straus Behavioral Research Facility.
- 11. At any point, if you decide that you want to seek treatment for your substance use, we will assist you in finding treatment.

#### WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

The risks and discomforts of this study are related primarily to the drugs given to you and the experimental procedures. We have carefully selected the doses to minimize the risk of serious side effects. Furthermore, some questions you will be asked throughout the study (about your medical, legal drug use history) may cause some discomfort.

The likely/most common risks of receiving opioid drugs include dizziness, stimulation, restlessness, a feeling of well-being, talkativeness, itchiness, nausea, vomiting, headache, constipation, dry mouth, sweating, sleepiness, light-headedness, and mild decreased breathing. These occasionally occur after receiving an opioid. These effects typically will go away on their own after a few hours and do not require any treatment. You should be familiar with these effects as you have used opioids previously. The risks of decreased breathing after administration of opioid drugs is related to the dose administered, and we have carefully selected doses to minimize the chance of serious decreases in breathing. If a serious decrease in breathing were to occur, this would be considered a very rare event that can be treated immediately and effectively with medication.

The likely risks of receiving alcohol include nausea, vomiting, headache, flushing, stimulation, sleepiness, drowsiness, feeling tired, changes in heart rate and blood pressure, changes in motor coordination, reaction time, vision, balance, hearing, and speech. These occasionally occur after receiving alcohol depending on the amount you use. These effects typically will go away on their own after a few hours and do not require any treatment.

We will watch you carefully throughout your participation to minimize the chance of any serious reactions.

We do not have any plans to draw your blood or conduct an electrocardiogram (ECG) after the screening is completed. However, if you were to get sick or hurt during the study, we may need to conduct these tests. There are risks related to drawing blood during screening or any time. Soreness, bruising, pain and a small amount of bleeding are likely to occur; fainting and infection are more rare. It is possible that we may have to try more than once to draw blood (which is not uncommon). An ECG is painless. Approximately 12 sticky pads will be placed on your skin and your heart's electrical activity will be measured. The electrodes may feel cold when first applied. In rare cases, some people may develop a rash or irritation where the patches were placed.

Exposure to drugs and alcohol may have harmful effects on a fetus or a newborn, and you will not be allowed to participate in the study if you are pregnant, planning to become pregnant or breastfeeding during the study, or if you cannot use an appropriate contraception method.

We will make every effort to keep private all research records that identify you to the extent allowed by law. However, there is a risk that a breach in confidentiality may occur. If this occurs, it may cause problems such as embarrassment and emotional stress.

There is always a chance that any medical treatment can harm you. The research medications and procedures in this study are no different. In addition to risks described in this consent, you may experience a previously unknown risk or side effect. We will do everything we can to keep you from being harmed.

#### WILL YOU BENEFIT FROM TAKING PART IN THIS STUDY?

You will not get any personal benefit from taking part in this study. However, if you take part in this study you may help us learn more about the effects of certain prescription opioids and alcohol when taken alone and together.

#### IF YOU DON'T WANT TO TAKE PART IN THE STUDY, ARE THERE OTHER CHOICES?

If you do not want to be in the study, there are no other choices except not to take part in the study. We can provide medical or drug treatment referrals to you if need them.

#### WHAT WILL IT COST YOU TO PARTICIPATE?

The study procedures and medications will be provided at no cost to you.

You and/or your insurance company, Medicare, or Medicaid will be responsible for the costs of all care and treatment that you would normally receive for any medical conditions you may have. These are costs that are considered medically necessary and will be part of the care you receive even if you do not take part in this study.

The University of Kentucky will not be allowed to bill your insurance company, Medicare, or Medicaid for the medical procedures done strictly for research.

## WHO WILL SEE THE INFORMATION THAT YOU GIVE?

We will make every effort to keep confidential all research records that identify you to the extent allowed by law. Your information will be combined with information from other people taking part in the study. When we write about the study to share it with other researchers, we will write about the combined information we have gathered. You will not be personally identified in these written materials. We may publish the results of this study; however, we will keep your name and other identifying information private. We will collect your social security number; this is required in order for you to participate.

We will make every effort to prevent anyone who is not on the research team from knowing that you gave us information, or what that information is. Your name will be kept separate from the information that you give, and these two things will be stored in different places under lock and key. Information collected electronically will be stored on password-protected computers.

You should know that there are some circumstances in which we may have to show your information to other people because we are required to.

For example, the law may require us to share your information with:

- a court or agencies, if you have a reportable disease/condition;
- authorities, if you report information about a child being abused; or if you pose a danger to yourself or someone else.

To ensure the study is conducted properly, officials of the Food and Drug Administration, the National Institutes of Health, the University of Kentucky, and the National Institute on Drug Abuse may look at or copy pertinent portions of records that identify you.

#### Certificates of Confidentiality (CoC):

To help us protection your privacy, this research has a Certificate of Confidentiality. The researchers can use this Certificate to refuse to disclose information that may identify you to anyone not connected with this study, or in any legal proceedings. The exceptions to this rule are release of information:

- you have requested us to provide, for instance, to your insurance company or doctor;
- to the sponsor (e.g., National Institutes of Health) or agency auditing the research (e.g., Food and Drug Administration);
- about child or elder abuse, neglect, or harm to yourself or others; and
- about you if it involves a reportable disease.

This policy does not prevent you from releasing information about your own participation in this study.

#### CAN YOU CHOOSE TO WITHDRAW FROM THE STUDY EARLY?

You can choose to leave the study at any time. You will not be treated differently if you decide to stop taking part in the study. If you choose to leave the study early, data collected until that point will remain in the study database and may not be removed.

The investigators conducting the study may need to remove you from the study. You may be removed from the study if:

- you are not able to follow the directions,
- we find that your participation in the study is more risk than benefit to you, or
- the agency paying for the study chooses to stop the study early for a number of scientific reasons.

If you stop the study because of side effects from the medication or another health-related reason, we will follow up with you by telephone or request that you come visit us so we can see how you are doing.

# ARE YOU PARTICIPATING, OR CAN YOU PARTICIPATE, IN ANOTHER RESEARCH STUDY AT THE SAME TIME AS PARTICIPATING IN THIS ONE?

You <u>may not</u> take part in this study if you are currently involved in another research study. It is important to let the investigator know if you are in another research study. You should discuss this with the investigator before you agree to participate in another research study while you are in this study.

#### WHAT HAPPENS IF YOU GET HURT OR SICK DURING THE STUDY?

If you believe you are hurt or if you get sick because of something that is due to the study, you should call Michelle Lofwall, MD, at **(859) 323-9321** immediately. Dr. Lofwall will determine what type of treatment, if any, is best for you at that time.

It is important for you to understand that the University of Kentucky does not have funds set aside to pay for the cost of any care or treatment that might be necessary because you get hurt or sick while taking part in this study. Also, the University of Kentucky will not pay for any wages you may lose if you are harmed by this study.

Medical costs related to your care and treatment because of study-related harm will be your responsibility.

You do not give up your legal rights by signing this form.

#### WILL YOU RECEIVE ANY REWARDS FOR TAKING PART IN THIS STUDY?

You will receive payment for taking part in this study. You will receive \$60 per night that you stay in the hospital. If you complete the study, you will receive an additional \$60 for every night of your stay (\$120/night if you complete). However, you will not receive this bonus if you are dismissed from the study, do not qualify after the qualification session is completed, or if you choose to quit the study before completion.

The total amount of money that you could earn by completing this study is approximately 3,600. This estimate is based on the average length of stay of 30 nights ( $120 \times 30$  inpatient nights = 3600); however, the number of days that you will stay may vary. This total does not include screening and follow-up payments.

You will also receive \$25 for your follow-up appointment scheduled approximately 2 weeks after your discharge from the study.

UK policy only permits us to pay participants in \$500 increments (meaning the maximum amount of each check is limited to \$500 per day). You will be given your first payment at discharge. We will mail you the remainder of the checks. We will mail you \$500 per check per day until you are fully paid. We will mail the checks to the address that you provide us or you can choose to pick them up in person if that is more convenient.

For example, if you complete the study and earn \$3,600, you will receive \$500 on the day of discharge and then will receive seven \$500 checks in the mail and a \$100 check in the mail  $(7 \times 500 + 100 = 3600)$ ; it will take approximately 2 weeks for you to receive all 8 checks. Alternatively, you are permitted to visit our office to pick up a check in-person during normal business hours Monday-Friday (closed on weekends, holidays).

Study payments are considered taxable income reportable to the Internal Revenue Service (IRS). You will be asked to complete a W-9 form which includes your name, address and Social Security number. A form 1099 will be sent to you if your total payments for research participation are \$600 or more in a calendar year.

# WHAT IF NEW INFORMATION IS LEARNED DURING THE STUDY THAT MIGHT AFFECT YOUR DECISION TO PARTICIPATE?

We will tell you if we learn new information that could change your mind about staying in the study. We may ask you to sign a new consent form if the information is provided to you after you have joined the study.

#### WILL YOU BE GIVEN INDIVIDUAL RESULTS FROM THE RESEARCH TESTS?

Generally, tests done for research purposes are not meant to provide clinical information. We will not provide you with individual research results.

### WILL WE CONTACT YOU WITH INFORMATION ABOUT PARTICIPATING IN FUTURE STUDIES?

The research staff would like to contact you in the future with information about participating in additional studies. If so, it will be limited to approximately 4 times per year.

| Do you give your permission to be contacted in the future by Dr. Walsh and/or the research team regarding |
|---|
| your willingness to participate in future research studies? |
| □ Yes □ No Initials |

#### WHAT ELSE DO YOU NEED TO KNOW?

This study is funded by the National Institute of Health/National Institute on Drug Abuse.

A description of this clinical trial will be available on www.ClinicalTrials.gov as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### WILL YOUR INFORMATION BE USED FOR FUTURE RESEARCH?

#### STORING AND SHARING YOUR INFORMATION FOR FUTURE USE:

The researchers would like to store, use, and share your identifiable information for future research use. Having information from many people helps researchers identify trends and discover better ways to diagnose, prevent, and treat many conditions. Researchers can use the stored information to learn more about substance use or research additional scientific questions.

#### WHERE WILL INFORMATION OR SPECIMEN SAMPLES BE STORED AND FOR HOW LONG?

The information will be stored at the Robert Straus Behavioral Research Facility for a minimum of 7 years.

# ARE THERE RISKS FROM ALLOWING YOUR INFORMATION OR SPECIMEN SAMPLES TO BE STORED FOR FUTURE RESEARCH?

There is a risk that someone could get access to the stored information or samples. In spite of the security measures and safeguards we will use, we cannot guarantee that your identity will never become known.

There may be risks that at this time are unknown. As technology advances, there may be new ways of linking information back to you that we cannot foresee now.

#### HOW WILL YOUR PRIVACY AND CONFIDENTIALITY BE PROTECTED?

Researchers will take careful steps to keep your information confidential.

Researchers will store your identifiable information, in a password-protected database to protect it from being accessed by anyone outside of the approved staff.

Researchers will remove your name or other direct identifiers from your information or samples. We will label your information or samples with a code and will store the key separately from the master code list. Only select staff will have access to the list that links the code to you.

# WHAT IF YOU CHANGE YOUR MIND AND WANT TO WITHDRAW YOUR INFORMATION OR SPECIMEN SAMPLES?

You may withdraw your permission to allow your information or samples to be used for future research. To do so, you must send a written withdraw request to:

Sharon L Walsh, Ph.D. 845 Angliana Ave Lexington, KY 40508

We will destroy any remaining information and samples that have been stored. In addition, it may be possible to destroy the code that links you with your information and specimen samples. However, we cannot withdraw the information and samples that have already been used.

#### WILL YOU RECEIVE ANY COMMERCIAL PROFIT FROM FUTURE RESEARCH DISCOVERIES?

The information and samples that you provide will no longer belong to you. The research may lead to new medical knowledge, tests, treatments, or products. These products could have some financial value. There are no plans to provide financial payment to you or your relatives should this occur.

#### WILL YOU BE GIVEN INDIVIDUAL RESULTS FROM THE FUTURE RESEARCH TESTS?

Tests done for research purposes are not meant to provide clinical information or help care for you. The results are only important for research. Therefore, the results of tests done with your information and samples will not be provided to you. In the rare event that a finding might affect the health of you or your family, we will contact you and you can choose whether to receive or refuse the information.

| <u> </u> |
|---|
| OPTIONAL FUTURE USE: |
| Do you give permission for Dr. Sharon Walsh to store your information for future research? |
| □ Yes □ No Initials |
| Remember, you can still be in the main study even if you even if you do not wish to allow your information stored for this investigator's future research. |

#### AUTHORIZATION TO USE OR DISCLOSE YOUR INDENTIFIABLE HEALTH INFORMATION

The privacy law, HIPAA (Health Insurance Portability and Accountability Act), requires researchers to protect your health information. The following sections of the form describe how researchers may use your health information.

### Your health information that may be accessed, used and/or released includes:

- Name and date of birth
- Demographic information (age, gender, ethnicity)
- Contact Information (street address, city or county of residence, email, phone number)
- · Social security number
- Results of physical exams, blood tests, ECGs, other diagnostic and medical procedures related to the study
- Personal medical history related to the study

### The Researchers may use and share your health information with:

- The University of Kentucky's Institutional Review Board/Office of Research Integrity
- Law enforcement agencies when required by law
- University of Kentucky representatives
- UK HealthCare and their representatives
- UK Health system (EPIC, the electronic medical records) and health systems outside of UK for which you
  have a patient relationship
- The U.S. Food and Drug Administration (FDA)
- The National Institute on Drug Abuse (NIDA)
- Investigational Drug Service (IDS) at the University of Kentucky
- Center for Clinical and Translational Science (CCTS) and Clinical Research Unit (CRU)

If you become pregnant anytime during the study or within 30 days after stopping the study drug, you must inform the study doctor. The study doctor must then report the outcome of your pregnancy to the Sponsor (and/or the FDA).

The researchers agree to only share your health information with the people listed in this document.

Should your health information be released to anyone that is not regulated by the privacy law, your health information may be shared with others without your permission; however, the use of your health information would still be regulated by applicable federal and state laws.

You may not be allowed to participate in the research study if you do not sign this form. If you decide not to sign this form, it will not affect your:

- Current or future healthcare at the University of Kentucky
- Current or future payments to the University of Kentucky
- Ability to enroll in any health plans (if applicable)
- Eligibility for benefits (if applicable)

# After signing the form, you can change your mind and NOT let the researcher(s) collect or release your health information (revoke the Authorization). If you revoke the authorization:

- Send a written letter to Dr. Sharon L. Walsh, to inform her of your decision. Her address is
  - Sharon L. Walsh. Ph.D.
  - 845 Angliana Ave
  - Lexington, KY 40508
- Researchers may use and release your health information already collected for this research study.
- Your protected health information may still be used and released should you have a bad reaction (adverse event).

You understand that you will not be allowed to review the information collected for this research study until after the study is completed. When the study is over, you will have the right to access the information. The use and sharing of your information has no time limit.

If you have not already received a copy of the Privacy Notice, you may request one. If you have any questions about your privacy rights, you should contact the University of Kentucky's Privacy Officer between the business hours of 8am and 5pm EST, Monday-Friday at (859) 323-1184.

# **APPENDIX – Detailed Study Calendar**

| | SCREENING | INPATIENT STUDY | | | | FOLLOW-UP |
|---|---|---|---|---|---|---|
| STUDY ACTIVITIES | 1-2 Weeks | Inpatient Week 1 | Inpatient Week 2 | Inpatient Week 3 | Inpatient Week 4 | 2-4 Weeks After<br>Study Completion |
| Informed Consent | • | | | | | |
| Urine/Breath Sample | • | | | | | |
| Labs/ECG | • | | | | | |
| Screening Questionnaires | • | | | | | |
| Physical Exam | • | | | | | |
| Questionnaires | | • | • | • | • | |
| Urine/Breath Samples | | • | • | • | • | |
| Study Sessions 1-3 times/week | | • | • | • | • | |
| Study Drug Administration | | • | • | • | • | |
| Session Questionnaires | | • | • | • | • | |
| Vitals/Safety monitoring | | • | • | • | • | |
| Brief Questionnaires | ì | | | | | • |

### **INFORMED CONSENT SIGNATURES**

This consent includes the following:

- Key Information Page
- Detailed Consent
- Appendix (Calendar)

You are the subject. You have read this information, and you will receive a copy of this form after it is signed.

| Signature of research subject | Date | |
|---|---|---|
| Printed name of research subject | | |
| Printed name of [authorized] person obtaining informed consent and HIPAA authorization | | Date |
| Signature of Principal Investigator or Sub/Co-Investigator | | |